# Title: Capnography-Assisted Learned Monitored (CALM) Breathing Therapy for COPD

Investigator: Annamaria Norweg, PhD

NCT04786184

**Unique Protocol ID: AAAT8556** 

**Protocol (Version August 22, 2022)** 

# RESEARCH STRATEGY

#### A. SIGNIFICANCE.

# A.1 Significance and Biological Relevance of the Proposed Clinical Trial.

Chronic obstructive pulmonary disease (COPD) is a leading cause of death and disability in the US and worldwide. <sup>1-3,4,5,6</sup> COPD is characterized by airway obstruction, hyperinflation, abnormal levels of carbon dioxide (CO<sub>2</sub>) and oxygen (O<sub>2</sub>), dysfunctional breathing patterns, and low physical activity (PA). Dyspnea (labored, uncomfortable breathing), the primary symptom of COPD, has devastating and debilitating effects on patients' physical and emotional well-being. <sup>7,8,9,10</sup> An estimated 15 million Americans (6.3% of the adult population) have COPD. <sup>11</sup> Its prevalence is increasing due to aging of the world's population, continued exposure to risk factors, and improved diagnosis. <sup>4,12</sup> There is a higher prevalence of anxiety disorders in COPD (up to ~50%) including panic disorder (PD; up to 10 times higher), than in the general population. <sup>13-15</sup>

**A.1.1 Dyspnea and Dysfunctional Breathing in COPD.** Dyspnea consists of several qualitatively distinct sensations, such as air hunger (a sense of insufficient air), increased "urge to breathe", "chest tightness", and feeling "starved for air". It relates to two main constructs: breathing effort and air hunger. Dyspnea is the principal reason that patients with COPD seek medical and rehabilitation services. Dyspnea is driven by chemosensors that sense abnormalities of CO<sub>2</sub> gases in the blood controlling inspiratory drive and mechanosensors in the ribcage (outside of the lungs) that sense the work of breathing. Dyspnea has sensory-perceptual (intensity and quality), affective distress, and impact or burden domains. Dyspnea and associated anxiety contribute to a vicious circle of abnormally rapid breathing (tachypnea), air trapping, and lung hyperinflation, leading to further dyspnea and PA limitations and impaired quality of life (QOL).

Dysfunctional breathing is "an alteration in the normal biomechanical patterns of breathing that result in intermittent or chronic symptoms". <sup>24,p.1-2</sup> People with COPD tend to breathe rapidly and shallowly through the mouth, relying on excessive upper chest and accessory respiratory muscle use, and hold their breath frequently. <sup>25</sup> This inefficient, thoracic-dominant breathing pattern (movement of upper thorax without lateral costal expansion<sup>26</sup>) contributes to dyspnea, CO<sub>2</sub> retention, and reduced exercise tolerance. <sup>27,28</sup> Both hypocapnia (low CO<sub>2</sub>) and hypercapnia (high CO<sub>2</sub>) occur in COPD depending on the stage of disease (**Fig. 2**). <sup>29,30</sup> Given that respiratory muscles are under both brainstem and skeletal muscle control, patients can learn self-regulated breathing to manage their symptoms. <sup>27,31-33</sup>

- **A.1.1.1 Low CO<sub>2</sub> Levels (Hypocapnia) and Dyspnea in COPD.** More than O<sub>2</sub>, abnormal CO<sub>2</sub> output is a marker of an inefficient breathing pattern. All patients with COPD demonstrate breathing inefficiency, marked by an elevated ratio of ventilation to CO<sub>2</sub> output (V<sub>E</sub>/VCO<sub>2</sub>). In mild to moderate COPD, fast breaths eliminate too much CO<sub>2</sub>, causing hypocapnia. Hypocapnia produces bronchoconstriction (airway smooth muscle contraction), bronchospasm, and vasoconstriction (decreasing pulmonary oxygen delivery), which reduce alveolar ventilation-perfusion matching (**Fig. 2**). Hyperventilation-induced hypocapnia creates an acid-base disturbance (alkalosis) inducing panic attacks. Emotions (stress, crying, and laughter), via autonomic vagal excitation, induce hypocapnia.
- **A.1.1.2 High CO<sub>2</sub> Levels (Hypercapnia) and Dyspnea in COPD.** In severe COPD, the pattern of breathing (abnormally rapid and shallow breaths) contributes to CO<sub>2</sub> retention (hypercapnia) (**Fig. 2**).<sup>45,46</sup> Hypercapnia then triggers anxiety and panic, especially in adults with anxiety disorders.<sup>47,48</sup> In a vicious cycle, rapid breathing due to exercise intolerance and emotional stress causes hypercapnia. Hypercapnia then increases ventilation, resulting in a cycle of increasing anxiety, panic, shortness of breath, and risk of ventilatory pump failure (neuromechanical dissociation), and related hospitalizations and mortality in COPD.<sup>49,50-52,53,54,49,55</sup> Chronic hypercapnia is associated with poorer prognosis in COPD.<sup>30</sup>
- **A.1.2 Anxiety, Abnormal CO<sub>2</sub>, and Impaired Interoception in COPD.** Anxiety in the sense of worry or nervousness is defined as "apprehensive anticipation of future danger" with both internal and external focus. <sup>56,p.7</sup> Panic is distinct from this more general anxiety or nervousness, because it relates to the feeling that a terrifying event is imminent or in progress <sup>56</sup> and can trigger an intense physical (e.g., dyspnea) and emotional response (e.g., extreme fear). Anxiety disorders include generalized anxiety disorder (GAD), PD, social anxiety disorder, and specific phobias. People with anxiety disorders also have elevated anxiety sensitivity (AS). <sup>57</sup> AS, a cross—anxiety disorder construct, is "the tendency of certain individuals to view interoceptive sensations as dangerous or threatening". <sup>58,p.384</sup> These distorted beliefs impair coping behavior and cause profound physiological dysregulation of respiration and autonomic nervous system. <sup>59</sup> High AS worsens anxiety and panic, particularly as patients become overly focused on and fearful of internal (interoceptive) sensations.

Common anxiety symptoms seen in people with COPD across anxiety disorders with high AS include respiratory dysregulation (i.e., hyperventilation, higher breathing variability, and sighing), ruminative flooding of thoughts, physiological hyperarousal, hypervigilance and attentional bias to threat, and profound avoidance of experiences associated with anxiety symptoms (e.g., avoiding dyspnea-causing activities). Anxiety increases inspiratory neural drive and is associated with overactivity of stress-related systems or excessive allostasis (adaptive processes of activating physiological systems to maintain homeostasis).

CO<sub>2</sub> hypersensitivity is considered a biological (neurochemical) marker of anxiety disorder.<sup>61</sup> Biomarkers are "traits that are specific to certain disorders or syndromes".<sup>66, p.322</sup> CO<sub>2</sub> challenges (inhaling air with greater proportion of CO<sub>2</sub>) have anxiogenic and panicogenic effects.<sup>61</sup> Greater anxiety and panic attacks are induced via CO<sub>2</sub> challenges (e.g., 5% CO<sub>2</sub> inhalation) in patients with anxiety disorders (especially those with PD) compared with healthy controls.<sup>61</sup> Panic attacks induced in the lab are associated with low CO<sub>2</sub> at end of exhalation or end-tidal (ETCO<sub>2</sub>) and high breathing variability.<sup>47</sup> Anxiety causes long-term changes in partial pressure of CO<sub>2</sub> (pCO<sub>2</sub>) related to accelerated and irregular breathing pattern.<sup>67</sup> Characteristic open-mouth breathing contributes to upper-chest, hypocapnic breathing, especially in anxious patients.<sup>39</sup> Patients with COPD and anxiety might have a lower set-point (neural coding) for CO<sub>2</sub> due to chemo-hypersensitization and greater sympathetic nervous system activation, subsequently increasing hyperventilation.<sup>36,38,68,69</sup>

Panic has been described as a "false suffocation alarm" in which patients show CO<sub>2</sub> hypersensitivity and abnormal pH buffering (an exaggerated compensatory alkalotic buffering) after hyperventilation and alkalosis.<sup>70</sup> Many of these panic-like features are present across anxiety disorders in patients who have high AS. Anxiety moderates the cerebral blood flow effect of CO<sub>2</sub> during hypocapnia and hypercapnia, explaining the greater symptoms of CO<sub>2</sub> changes with anxiety disorders (**Fig 2**). Anxiety results in extreme awareness of interoceptive sensations, causing lower accuracy of signals.<sup>71,72,62</sup> Lower accuracy is experienced as distorted or amplified dyspnea disproportionate to lung function.<sup>73</sup>

#### A.1.3 CALM Breathing.

**A.1.3.1 CALM Breathing Core Exercises and Components.** CALM Breathing is a 4-week complementary, mind–body breathing therapy with biofeedback. It links CO<sub>2</sub> changes to dyspnea and anxiety symptoms and targets breathing efficiency and self-efficacy in COPD. It addresses dysregulated, inefficient breathing patterns (habits) and faulty beliefs or interpretations of dyspnea symptoms as key modifiable determinants of abnormal CO<sub>2</sub> levels and poor symptom management.<sup>25,26</sup> CALM Breathing focuses on helping participants to regain quicker breathing control and recovery when challenged to reduce dyspnea distress.<sup>74</sup>

CALM Breathing consists of eight 1-hour sessions, twice per week, and 10 core exercises, which are all guided by capnography biofeedback (**Table 1**). Each core exercise is followed by a debriefing to explore participants' responses and discuss related beliefs and any misconceptions. An example of a misconception is that dyspnea indicates that one needs more air.<sup>75</sup> Participants learn to identify dyspnea contextual cues and triggers (conditioned stimuli) and reinforcements to unlearn dysregulated breathing pattern habits.<sup>76,77,78</sup> During debriefings, the interventionists monitor any relaxation-induced anxiety (RIA) to help prevent it leading to panic. RIA is "paradoxical increase in physiological, behavioral, and cognitive aspects of anxiety with efforts to relax".<sup>79,p,2</sup> Participants are asked if they became more tense or experienced any disturbing or worrisome thoughts, memories, or images.<sup>80</sup> RIA can be overcome during slow breathing therapy.<sup>79</sup>

Fundamental to CALM Breathing is the application of motivational interviewing (MI) principles to establish a collaborative relationship and cultivate change talk.<sup>81</sup> MI is a "client-centered counseling style for eliciting behavior change by helping clients to explore and resolve ambivalence".<sup>82,p.326</sup> In each session, collaborative goals are set for home-based exercises for three target behaviors: 1) slow breathing pattern, 2) completion of home breathing exercises, and 3) lifestyle physical activity perseverance.<sup>83</sup>

**A.1.3.2 CALM Breathing: Capnography Biofeedback.** Biofeedback is a coaching, behavioral method that offers continuous, live feedback of physiology. <sup>84,85</sup> Capnography works synergistically with breathing therapy. Capnography measures and records pCO<sub>2</sub> in exhaled breath (ETCO<sub>2</sub>), which is a measure of pulmonary gas exchange. <sup>35,86</sup> A capnograph offers both numeric values of CO<sub>2</sub> and qualitative information on airflow patterns (e.g., breath holds or apneas, <sup>87</sup> sighs, effort, aborted exhales, and breath-to-breath regularity). <sup>88,87</sup> Exhaled CO<sub>2</sub> also provides a reliable measurement of RR. <sup>89</sup> Objective biofeedback data of ETCO<sub>2</sub>, RR, and airflow patterns in CALM Breathing provide clear, immediate biofeedback to guide breathing therapy.

The primary study capnograph will be the FDA-approved Handheld Capnograph and Oximeter (PC-900B, CMI Health, GA) in-session, with integrated arterial oxygen saturation (SpO<sub>2</sub>) sensor (**Fig. 1A**). The accuracy

of the Capnograph is ±2 mmHg for values of 0–40 mmHg and ±5% for values >41–70 mmHg, which meets International Organization of Standardization (ISO) standards for CO<sub>2</sub> reading.<sup>90</sup> The Capnograph will be used with nasal cannula. We will also use the CapnoTrainer<sup>91</sup> to display CO<sub>2</sub> waveforms in-session (**Fig. 1B**).<sup>89</sup>

| Tab | e 1. CALM Brea | thing Core Exercises. |
|---|---|---|
| | Exercise | Description |
| 1. | Slow, nasal respiration Exercises are quiet, nasal inhalation and exhalation (≤10−12 breaths per min at rest) <sup>92,93</sup> focused on lengthening exhalation. Practice is predominately relaxed (eupneic) breathing in supine as well as in sitting and standing recovery postures (e.g., supine or semi-recline positions, forward-leaning in standing or sitting with hands supported). <sup>77,94,95</sup> In later sessi slow breathing is practiced with tailored, simulated breathing challenges (e.g., speaking free walking and talking, or timed mental arithmetic) for transfer of learning. <sup>96</sup> | |
| 2. | Pursed-lips<br>breathing<br>(PLB) | PLB is "nasal inspiration followed by exhalation through partially (almost) closed [relaxed] lips,"97,p.344 focused on lengthening exhalation, with tailored ≤ 5-min physical challenges, chosen by participants (e.g., stepping in place, walking, or stair-climbing).77 |
| 3. | Positioning of the tongue | Participants practice placing and maintaining their tongue on the roof of their mouth (behind top teeth on hard palate) to correct open mouth breathing and facilitate nasal breathing with closed lips. Open-mouth breathing impairs respiratory mechanics and exercise tolerance, contributes to forward head posture, and is a risk factor for obstructive sleep apnea. <sup>98,99</sup> |
| 4. | Control pause (CP) | CP is a breathing maneuver post-exhalation of ~2–5 seconds; participants notice and count the length of the natural pause between breaths. Increasing pause time is important to slow the breath. Exercise facilitates regaining trust in the body's physiology. The three phases of the breath are emphasized: 1) inspiration, 2) post-inspiration, and 3) expiration (pause). 100,101 |
| 5. | Volume-<br>regulation | Exercises focus on regulating size and/or depth of breaths (or breath volume) for more efficient breathing (less wasted ventilation). <sup>27</sup> |
| 6. | Breathing interoceptive awareness | Width breathing: Participants notice and allow their lower ribs to laterally expand and elevate sideways and contract (bucket-handle motion). Length breathing: Participants feel their belly rising and falling, and ribcage elevating and lowering (pump-handle motion). Patients learn to de-recruit abdominal expiratory muscles for energy efficiency. Sighing is discouraged because it triggers arousal. Exercises facilitate allowing rather than habitual manipulating of the breath. |
| 7. | Breath<br>counting | To promote slow breathing and improved interoceptive accuracy ("objective accuracy to detect bodily sensations"), 104,p.130 participants count breaths in sets of 5–10 breath counts (e.g., "in, out, pause, 1; in, out, pause, 2" and so on) initially cued by the therapist and then practiced independently. |
| 8. | Humming | Humming is a type of resistance breathing pattern used to promote rhythmical, prolonged exhalation cued with participants' preferred music. <sup>105</sup> |
| 9. | Breathing<br>differentiation<br>training | Biofeedback facilitates differentiating rhythmical versus arrhythmic breathing (e.g., breath-holds, aborted breaths, avoiding transition times) to facilitate interoceptive accuracy. <sup>48</sup> Participants learn to estimate their ETCO <sub>2</sub> levels and accurately count their number of breaths based on interoceptive cues. They learn to differentiate somatic cues and ETCO <sub>2</sub> changes resulting from breathing (e.g., shallow versus deeper breaths). |
| 10. | Coordinated breathing | The exhalation phase of the breath is coordinated with ribcage stretches. 106 Breathing exercises with movement improve body awareness, grounding (reconnection with the body), 107 and sense of embodied self; 108 relieve muscle tension; and improve chest wall mechanics. Ribcage stretches include active shoulder rolls, head rolls, arm reaches overhead, forward bends and spinal rolls, pelvic tilts, side bends, spinal twists, and thoracic extensions. |



Figure 1. A) Capnograph PC-900B; B) CapnoTrainer, including capnogram. C) MightySat™ pulse oximeter with RR biofeedback.

**A.1.3.3 CALM Breathing Home-Based Exercises and Adherence Strategies.** Participants will be encouraged to practice home breathing exercises (especially audio-guided *slow nasal respiration* and *coordinated breathing* with RR biofeedback) for 10–20 min per day. Participants will receive a printed-out

"Home Breathing Exercises" hand-out during their first session. In addition, PLB with physical exertion will be promoted. Adherence strategies include collaboratively setting goals (action plans), logging home breathing exercises for self-monitoring, and therapist monitoring of recorded RR data. 109,110,83,111 At home, participants will use the MightySat<sup>TM</sup> fingertip pulse oximeter device for RR biofeedback to monitor their slow breathing exercises (**Fig. 1C**). Participants will receive a printed out "Pulse Oximeter" education hand-out during their first session. The FDA-approved RR biofeedback device uses photoplethysmography and algorithms to detect variations in blood flow and volume in skin; accuracy is verified for 4–70 bpm. 112-114 MightySat device uses Bluetooth to interface with a health app and stores 72 hours of data. Participants will be trained to use the MightySat<sup>TM</sup> in the first CALM Breathing session; its correct use will continue to be reinforced in-session (to ensure safety and quality of home practice).



Figure 2. CALM Breathing Conceptual Model.

**A.1.3.4 CALM Breathing: Conceptual Framework.** *Generative Model of Perception.* <sup>48</sup> This is a top-down neuropsychobehavioral model based on recent understanding of normal brain functions involved in the perception of bodily sensations. The brain represents the world by both exteroceptive sensations (e.g., sight) as well as interoceptive sensations from inside the body. Interoception is "the sense of the internal physiological condition of the body"<sup>115,p.971</sup> monitored by the nervous system for survival and evolutionary adaptation to the environment. <sup>17,65</sup> It is the mind's way of listening to the body. Interoception consists of monitoring of blood chemistry (CO<sub>2</sub>), afferent sensory stimuli from visceral organs, and interoceptive perceptions and inferences. <sup>115</sup> Breathing is one of several interoceptive channels. <sup>65</sup> The brain is continuously generating, testing, and reforming predictions ("best guesses") based on sensory data and prior expectations. <sup>116</sup> The brain learns to minimize differences between predictions and sensory signals (prediction errors or surprise) and optimize homeostatic-allostatic control via autonomic reflexes as a regulator for survival. <sup>48</sup> When sensory inputs are noisy and unclear (have low inferred precision), which is common with anxiety, interpreting internal states is influenced by priors (reducing influence of sensory inputs). <sup>117</sup> Priors are cognitions and emotions that actively contribute to perception. Stress symptoms stem from low allostatic self-efficacy (a metacognitive belief of low capacity to self-regulate bodily states, such as dyspnea).

*Interoceptive Exposure and Learning Theory*. <sup>56,118</sup> Through interoceptive exposure to breathing sensations, CALM Breathing is theorized to reduce CO<sub>2</sub> hypersensitivity and physiological arousal to respiratory stimuli. <sup>60,72,119,120,73</sup> Exposure to breathing stimuli without negative consequences is designed to extinguish

classically conditioned emotional responses to breathing stimuli.<sup>56,60</sup> The rewards of more regulated breathing are reinforced. Interoceptive exposure promotes subjective sense of physiological well-being and trust of the body.<sup>60,121</sup>

**A.1.4 Knowledge Gaps.** COPD clinical studies have not adequately focused on breathing therapy that includes anxiety and physiological measures as important endpoints. <sup>122, 123, 33</sup> While breathing strategies are strongly supported for dyspnea relief and exercise tolerance by expert opinion, existing evidence is from small-scale studies. <sup>77</sup> PR is a comprehensive intervention that includes aerobic and strengthening exercise training, breathing exercises, and education. <sup>77</sup> While PR is effective in improving dyspnea, QOL, and exercise capacity in COPD, <sup>124</sup> the contributions of breathing therapy exercises, a component of PR, are less known. Anxiety is associated with worse PR outcomes: greater dyspnea and perceived functional impairment post-PR, and worse QOL and 6-minute walk distance (6MWD). <sup>125,126</sup> Therefore, there are knowledge gaps for how to improve PR outcomes, including uptake, especially for anxious patients. <sup>127</sup>

**A.1.5 Barriers and Treatment Limitations in Symptom Management for COPD.** Currently there are limited dyspnea and anxiety treatment options, and management is suboptimal.  $^{128,129,70,130}$  The standard of care for COPD is pharmacotherapy and supplemental  $O_2$ ,  $^{12}$  but bronchodilators and corticosteroids provide only minor relief of dyspnea and airflow obstruction.  $^{19,38}$  Supplemental  $O_2$  relieves dyspnea by slowing breathing pattern and reducing hyperinflation.  $^{131}$  However, short-term supplemental  $O_2$  use has low patient acceptability.  $^{132}$ 

Because a comprehensive PR program can improve symptoms, exercise tolerance, and QOL, guidelines strongly recommend it, but it is grossly inaccessible to most patients with chronic lung diseases and underutilized worldwide. 127,133,134 Overall real-world uptake of PR by patients with COPD is 1–2% due to significant barriers. 135 A recent systematic review identified key barriers to PR uptake in COPD as fear of dyspnea, fear of exercise and exhaustion, and belief it would not be beneficial, among other reasons. 136 Recent studies further suggest that PR post-acute exacerbation of COPD (AECOPD) might not be acceptable for patients, with an uptake of only 9%. 137,138,139 Based on our research, real-world PR drop-out rates in COPD are >40%. In one study (N = 128), the main reason for not attending an initial PR assessment or dropping out post-AECOPD was feeling unwell or too breathless. 137 PR teaches pursed-lips breathing only during physical exercise challenges, when a person's respiratory system and emotional state are typically significantly stressed, and mechanical and chemical demands are greatly amplified, possibly limiting the opportunity to learn self-regulated breathing. By not addressing anxiety, PR offers more limited learning opportunities for desensitization, and exposure to dyspnea in PR may actually trigger increased anxiety in some anxious patients. Therefore, PR doesn't address breathing irregularity and anxiety simultaneously, which is essential to optimizing treatment in COPD. 140 In contrast, CALM Breathing is designed to extinguish emotional responses to breathing mechanics and CO<sub>2</sub> symptoms.

Inspiratory muscle training using devices that add a resistive load to strengthen inspiratory muscles does not improve COPD clinical outcomes.<sup>77,141</sup> In addition, noninvasive positive pressure ventilation (NPPV) might be a useful adjunct to PR for COPD to unload respiratory muscles to relieve dyspnea.<sup>77</sup> However, NPPV is a labor-intensive, costly intervention, requiring expertise to use it, and has low adherence and high drop-out rates (up to 44%) because of discomfort.<sup>142</sup> NPPV might not be practical in a non-hospital setting.<sup>142</sup>

The efficacy of traditional cognitive-behavioral therapy (CBT) treatments for anxiety and dyspnea in COPD is uncertain. CBT compared with a control condition in a meta-analysis had only a small effect on improving anxiety in older adults, indicating a need for new approaches. Adults with hypocapnia were twice as likely to drop out of CBT. A meta-analysis found low quality evidence of the efficacy of psychological therapies for COPD and anxiety. Breathing retraining is not offered to patients with COPD outside of rehabilitation.

Breath practices are also central to yoga, tai chi, and other Eastern traditions. While a few studies are underway or have been completed, 149-153 scientific evidence of their efficacy as adjunctive treatments in PR is still very limited. 154, 155 Further, limited data is available outside Asian populations. 146 Evidence to date suggests these therapies may not be fully accepted by Western populations with COPD; for example, in a mindfulness study of men with moderate to severe COPD, 52% of participants withdrew. 156 Further, yoga in its many forms may also need to be adapted to better target the breathing challenges of COPD for optimal benefit. More than increasing interoceptive awareness, with scientific premise, CALM Breathing systematically targets dysfunctional breathing patterns to promote slow, eucapnic breathing and interoceptive breathing accuracy and self-efficacy specifically for dyspnea symptom relief. 99

A critical barrier to progress in the field of anxiety management for COPD is stigma associated with the classification of anxiety as a mental illness.<sup>13</sup> Many patients with COPD delay seeking treatment for anxiety or go without needed care. CALM Breathing might be a more acceptable, less stigmatizing mind–body intervention compared with traditional mental health interventions,<sup>147</sup> and may improve anxiety and dyspnea.

There is little and conflicting evidence for the use of antidepressant and anxiolytic medications for relieving dyspnea and improving QOL.<sup>130</sup> Psychopharmacological treatments for anxiety have reduced long-term efficacy and can cause severe side effects, dependence, adverse reactions, cognitive impairment, and falls, as well as addiction and relapse in older adults.<sup>70,130,148-151</sup> Medication does not build long-term coping and information-processing skills or behavior change.<sup>107</sup> International practice guidelines recommend an integrative approach of combining medication with psychological or mind–body interventions.<sup>12,152</sup>

**A.1.6 Significance and Impact of the Study in Clinical Practice.** This trial addresses two significant comorbidities, anxiety and COPD. The gained knowledge could change the treatment paradigm for COPD patients. <sup>127,153</sup> CALM Breathing has potential important downstream effects on reducing fearful activity avoidance. ETCO<sub>2</sub> biofeedback simplifies learning to promote breathing and PA behavior change. <sup>154</sup> CALM Breathing focuses on reducing dyspnea and safety-seeking behaviors that contribute to deconditioning, a sedentary lifestyle, and persistence of a cycle of high anxiety levels. Compared to traditional PR, the monitored home-based breathing exercise program boosts therapy dose, and establishes routines for long-term behavior change. <sup>153,110,155</sup> This study addresses a critical knowledge gap of how to improve PR use. CALM Breathing offers a needed bridge or stepping-stone to prepare patients for PR to potentially improve PR utilization. <sup>12,136,156,157,138,156</sup> As such, CALM Breathing meets the definition of a *transitional care intervention* ("a time-limited intervention designated to promote safety and timely transfer of patients across care settings" <sup>158</sup>).

Expert consensus supports establishing *breathlessness rehabilitation* for COPD.<sup>153</sup> In a recent breathlessness workshop for COPD and chronic heart failure with 74 stakeholders, only 36% agreed with the statement "exercise training was the most important component of rehabilitation for breathlessness".<sup>153,p. 235</sup> Instead, they believed that psychological and educational components of rehabilitation were also important for dyspnea remediation.<sup>153</sup> As advocated by these stakeholders, by preceding exercise training, CALM Breathing may work in synergy with PR to improve physical and mental health outcomes.

#### B. INNOVATION AND GENERALIZABILITY OF POTENTIAL FINDINGS.

CALM Breathing, a complementary approach and adjunct to PR, is innovative because:

- i. Novel therapeutic targets of ETCO<sub>2</sub> and RR levels are used to improve both breathing pattern efficiency and anxiety in COPD; immediate goal-directed feedback of capnography nudges skill acquisition.<sup>78,140,94,88,89</sup> CALM Breathing uses a novel application of capnography to integrate CO<sub>2</sub> biofeedback with breathing therapy while attending to anxiety sensitivity.<sup>159,160</sup>
- ii. Timing of CALM Breathing (before PR) offers a phased approach to PR uptake to address important barriers to PR acceptance, readiness, and utilization.
- iii. CALM Breathing includes novel home-based device-assisted RR biofeedback and data recording to monitor breathing exercise quality, motivate behavior change, and enable adherence checks. 153,110,155
- iv. Our approach includes novel physiological and anxiety outcome measures, including change in ventilation patterns (RR and ETCO<sub>2</sub>), lacking in other COPD breathing therapy studies.
- v. Innovative coaching (MI) is implemented, which emphasizes collaboration and shared decision making.
- vi. CALM Breathing translates neuroscientific understanding of sensory perception to treat dyspnea. 48,161

CALM Breathing is scalable because it does not rely on smartphone delivery. This could be important for older patients, as the use of smartphones in adults 65+ years old is only ~53%. 162

# C. SUPPORTING DATA, CLINICAL EVIDENCE, AND RATIONALE FOR THE PROPOSED CLINICAL TRIAL.

#### C.1 Benefits of Slow Breathing.

Slow breathing activates the parasympathetic nervous system, via the right and left vagus nerves, to soothe and calm the mind. Slower RR prevents a feedback cycle of panic in a dyspnea crisis to prevent ventilatory pump failure. Slow PLB reduces anatomical dead space (V<sub>D</sub>) and increases the amount of CO<sub>2</sub> removed (breathing efficiency) as its primary mechanisms in COPD. He reduces hypercapnia by improving the elimination of CO<sub>2</sub> and alveolar-capillary diffusion. L4,165-167 PLB decreased ETCO<sub>2</sub> and RR in patients with

severe COPD.<sup>168</sup> PLB has been endorsed in evidence-based practice guidelines to relieve dyspnea in advanced COPD.<sup>128,130</sup> PLB reduced RR and increased tidal volume in a systematic review.<sup>169</sup>

Device-guided slow breathing training when combined with PR program (using a pneumotachometer interfaced with a computer display of respiratory and goal feedback) reduced dynamic hyperinflation in moderate to severe COPD compared with both PR alone and breathing training alone.<sup>32</sup> Adherence was 75–76.5% for research-based PR. Both ventilation feedback groups slowed their breathing by increasing expiratory time, supporting the benefits of goal-directed biofeedback in breathing therapy.

# C.2 Device-Guided Capnometry-Assisted Respiratory Training (CART) Approach.

Participants with PD (N = 69) receiving a 4-week capnometry-guided respiratory intervention had improved panic severity, increased ETCO<sub>2</sub>, and improved anxiety control.<sup>170</sup> Also, CART increased ETCO<sub>2</sub>, decreased distress, and improved asthma symptoms at follow-up in adults with asthma compared with a comparison group of slow breathing and awareness training (SLOW) with RR feedback alone (N = 120).<sup>31</sup>

## C.3 Role of Recovery Postures and Chest Wall Stretches with Breathing Exercises in COPD.

For hypercapnia, the energy demands of breathing are reduced by supine and forward-leaning postures with arms supported. Supine posture augments prolonged expiratory time and abdominal ribcage tidal volume compared to sitting (p < 0.01). In a study (N = 23), 13 adults with COPD showed paradoxical indrawing movement of the lower ribcage with inspiration in sitting, which was corrected by a supine posture. Recovery postures allow cephalad positioning of the diaphragm and ribcage, reduce a kyphotic posture, improve chest wall compliance for improved efficiency of the ventilatory pump, and regulate autonomic nervous system arousal. Chest wall muscle stretches and augmentative postures inhibit activation of accessory muscles of respiration and facilitate synchronous motion of the chest and abdomen.

## C.4 Relationship between ETCO<sub>2</sub> and PaCO<sub>2</sub>.

ETCO<sub>2</sub> is a good estimate of arterial pCO<sub>2</sub> for patients with stable COPD in non-acute respiratory distress and spontaneously breathing (non-intubated) (r = 0.89). The end of the end

#### D. APPROACH.

### D.1 Supporting, Preliminary Data from Research Team.

This study builds on our previous pilot trial called Capnography-Assisted Training in COPD to slow the BreatH (CATCH) (N=31).<sup>176</sup> CART was combined with a 10-week PR program. Randomization to CART+PR or PR alone was 2:1. Thirty-one participants with mild to very severe COPD enrolled in the study; 58.1% were female; 32.2% had mild to severe GAD-7 anxiety symptoms; and 30.8% were taking anxiety or depression medication. Adherence to CART sessions was 73.5% overall (n=22) and 100% for participants who completed PR (n=13). CART participants completed 61% of home breathing exercises based on logs. Mean number of PR sessions completed was 14.14 (7.37) for CART+PR and 11.44 (9.81) for PR alone (n=31). Fourteen people with mild to very severe COPD were also interviewed post-treatment using a topic guide. The identified five main themes: *PR Adherence*, *Learning to Breathe*, *Impact on Health*, *CART Dose*, *Recommending CART to Others* (Table 2). A majority (67%) of participants requested more than six CART sessions for maximum benefit. Results provided preliminary evidence of the feasibility and acceptability of CALM Breathing exercises, session structure and therapy space needed, and coaching approach (MI). Participants' feedback was used to refine CALM Breathing (e.g., frequency, timing, session structure, and home-based breathing exercises). For example, we simplified the home breathing exercises and biofeedback device, revised symptom tracking, and added written goals and confidence ruler to the exercise log. 159,111 We also revised the interview questions.

| Table 2. Example Themes and Quotes of Acceptability of CART- CATCH Study. | | |
|---|---|---|
| Theme | Subthemes | |
| Adherence | | It helped me to get along with and keep up and not give up. (ID: 1016, Female, 75 yrs) |
| Learning<br>to Breathe | CO <sub>2</sub><br>Biofeedback | The one thing I really enjoyed was the capnometer and seeing the breaths. Seeing a physical measure of what a breath is As soon as I saw what a good breath was, and what bad breathing was, on the moving graph then it kind of reinforced the way I should be breathing. (ID:1008, Male, 78 years) |

| | Mind–Body<br>Connection | The fact that I have been able to see on the screen the difference in being able to relax, focus on my breathing, the intake of air and exhalation, and seeing it on the screen and the differences. I saw a big difference and not only do I see it, but I feel itI've been aware of how my feelings impact my breathing andhow I can regulate and change it and I think that has been extraordinarily helpful. (ID: 1025, Female, 82 years) |
|---|---|---|
| Impact on | Relief of | I felt like it helped a lot because I've become aware of my breathing and I think I was |
| Health | Dyspnea | breathing much more shallowly before. I would always hold my breath on exertion, so it |
| | | basically, solved a lot I didn't realize that I was breathing the way I was I don't think I |
| | | was breathing as regularly or as in control as I am now. (ID: 1024, Female, 75) |
| | Reduced | It helped not only with the breathing itself, but even with the calming of the nerves |
| | Anxiety | Especially people that are nervous about it, just controlling your breathing, you automatically calm down. (ID: 1011, Female, 61 years). |
| | | It's like all stops because you are concentrating on [breathing], and it's peaceful there. So, I really liked that part. It stays with you. Because you know, if you can be calm and you can be peaceful, you can be breathing all right. And you won't be feeling those frightening feelings. (ID: 1030, Female, 65 years). |

In our observational study (N = 445) of adults with COPD, 36% of participants had mild to severe GAD-7 anxiety symptoms. We found self-reported physician diagnosis of anxiety even higher with a prevalence of  $42\%.^{140}$  In our study on anxiety and COPD (N = 182, mean age  $52 \pm 16$  years),  $^{57}$  50% had any of six anxiety disorders with a DSM-IV-based screening. A higher Anxiety Sensitivity Index (ASI) score was independently associated with higher dyspnea severity, more activity avoidance due to dyspnea with obstructive lung disease, and poorer ratings of subjective health.  $^{57}$  Mean ASI score was 18.4 for those with dyspnea.

#### D.2 Recruitment and Clinical Trial Experience.

Our study team has successfully collaborated on previous COPD and breathing therapy research.<sup>176,177</sup> Dr. Norweg has successfully recruited over 600 patients with COPD in her research work. Our team also has an extensive track record of publishing our clinical trials.<sup>176,178-180</sup>

#### D.3 Experimental Approach.

- **Aim 1:** To evaluate the feasibility of CALM Breathing before PR.
- **Aim 2:** To measure the acceptability of CALM Breathing before PR.
- **D.3.1 Study Design.** To achieve Aims 1 and 2, we will use a single-blind prospective RCT. In Phase I, participants will be randomized 1:1 to one of two groups: CALM Breathing (N = 20) and Wait-List control (N = 20). In Phase II, both groups will be offered a 10-week PR program (care as usual). Access to timely initiation of PR will be facilitated. We will use a hybrid design to evaluate feasibility and acceptability.<sup>181</sup>
- **D.3.1.1 Rationale for Study Design.** Why Use a Waitlist Design? We chose a waitlist control group as a usual care comparison group because PR intake evaluations are typically scheduled 6 weeks in advance of implementation. Therefore, 4-week CALM Breathing could fit seamlessly into PR programs and not delay standard of care. A qualitative study found that waiting for PR increased patients' feelings of uncertainty and lack of control regarding their care. Sour experience shows that once referred to PR, patients are motivated to start some form of therapy right away. CALM Breathing can leverage patients' motivation and reduce feelings of uncertainty. A target sample size of 40 subjects is justified based on the primary outcomes of feasibility and acceptability, and transition of participants to a 10-week PR program.
- **D.3.1.2 Rationale for Study Need.** This study is part of our phased approach to refine, optimize, and test the feasibility of CALM Breathing. Preliminary participant feedback from our CATCH study was applied to adapt and design CALM Breathing (including its dose, schedule, delivery, and home program). This pilot builds on initial lessons learned and identifies intervention areas still needing greater development to assure the success of a future large trial, targeting a subpopulation at risk, that is, those with COPD and anxiety.

The purpose of this pilot study is to establish success benchmarks of CALM Breathing and to test feasibility of:

- 1) recruiting a target group of adults with COPD and concurrent anxiety, including building a partnership with Columbia University Irving Medical Center's (CUIMC's) pulmonary department; ensuring adequacy of recruitment and study referral procedures;
- 2) using ASI-16, DMQ-CAT, and VAS dyspnea anxiety assessments for eligibility screening;
- 3) randomizing participants to CALM Breathing and Wait-List;

- 4) assessment procedures; confirming our estimates of time needed to administer assessments; evaluating participant ratings of assessment burden; and testing that target timelines and blinding are achievable; 183
- 5) facilitating timely PR intake assessment initiation (to limit wait);
- 6) implementing manualized CALM Breathing, including adequacy of dose (timing, frequency, and session duration), fidelity procedures, and transportation funds; attention will be given to additional considerations and tailoring needs of patients with significant anxiety sensitivity and/or anxiety disorders;
- 7) implementing home-based breathing exercise component (e.g., new RR device fidelity checks and new distribution of therapist-guided audio exercises using an MP3 player to improve adherence rate);<sup>181,184,185</sup>
- 8) retaining participants at 3-month follow-up post-PR, including ensuring adequacy of retention strategies.
- D.3.2 Participant Eligibility and Recruitment. Participants will be recruited from CUIMC's / New-York Presbyterian Hospital's outpatient PR program patient referral list. Participants will also be recruited from a cooperating clinical site, CUIMC's / New-York Presbyterian Hospital's Pulmonology Medicine Department, CUIMC'S/ New-York Presbyterian Hospital's Primary Care Medicine Department and New-York Presbyterian Lawrence Hospital Pulmonology Medicine Department. We will also plan to make use of CUIMC's RecruitMe platform. To facilitate participant recruitment and partnership building, we will partner with the Dr. Angela DiMango, MD and Dr. Charles Murphy, MD from CUIMC's/New-York Presbyterian Hospital's Pulmonology Medicine Department and Dr. David Buchholz from CUIMC's/New-York Presbyterian Hospital's Primary Care Medicine Department. CUIMC has a high volume of racially diverse patients with COPD. Feasibility of conducting this study is facilitated by a single Institutional Review Board (IRB) and a single-clinic recruitment site.
- **D.3.2.1** *Inclusion Criteria*: Eligible participants will be adult males or females with COPD in stable condition; have elevated anxiety symptoms; <sup>57,186</sup> have dyspnea symptoms; and require ≤8 hours per day of supplemental oxygen. All participants will receive standard care of pharmacotherapy with bronchodilators. <sup>77,12</sup> Participants taking anti-anxiety medication (e.g., selective serotonin reuptake inhibitors, SSRIs, and serotonin norepinephrine reuptake inhibitors, SNRIs) must be stably medicated for at least 4 weeks prior to study entry, <sup>152</sup> with no plans to change psychotropic medication dose.
- **D.3.2.2 Exclusion Criteria**: Participants may not have suicidal ideation or suicidal behaviors within the past year (score of >1 on psychologist interview-administered Clinician Suicide Assessment Checklist, which is a Modified Columbia-Suicide Severity Rating Scale-CSSRS). Participants cannot have morbid obesity (body mass index (BMI) > 40) or neuromuscular disease or be pregnant. Participants not eligible for CUIMC's PR program and those who have received PR training in past 12 months will be excluded. Concurrent receipt of short-term or new physical therapy, speech therapy, mindfulness, or meditation-based therapies (e.g., Mindfulness Based Stress Reduction) will not be permitted. Cognitive impairment will be screened by the Mini Mental State Exam, with score of ≤23 used as an exclusion criterion, to control for cognitive impairment and learning challenges. See Study Record for full eligibility criteria.
- **D.3.2.3 Rationale for Eligibility Criteria.** Assessments for elevated anxiety symptoms are based on our previous research. <sup>22,57,189</sup> No diagnosis of an anxiety disorder is required since participants with elevated anxiety symptoms could benefit from CALM Breathing. An inclusion criteria of anxiety symptoms (rather than anxiety disorder) increases the generalizability and potential impact of CALM Breathing, targeting anxiety and somatic symptoms such as occur with breathing in COPD. We will use accepted standards of spirometry testing to classify COPD patients (using grades 1 to 4) according to severity of airflow limitation. <sup>12</sup> Neuromuscular disease can affect PaCO<sub>2</sub>. <sup>30</sup> Obesity is associated with hypercapnia. Our threshold of hypercapnia of ETCO<sub>2</sub> > 50 mmHg is widely used. <sup>190</sup> Pregnancy can reduce ventilatory control, resulting in hyperventilation, hypocapnia, and alkalosis. <sup>191</sup> We have attended to prescription medication as a confounder. We will adjust for stable antidepressant use (SSRIs and SNRIs) in statistical analyses. Excluding patients taking antidepressants would reduce generalizability. <sup>192</sup>

#### D.3.3 Study Groups and Interventions.

- **D.3.3.1 Capnography-Assisted Learned, Monitored Breathing (CALM) Intervention.** The 4-week CALM Breathing therapy will consist of eight 1-hour individual treatment sessions over 4 weeks pre-PR (**Tables 1, 3–4** and section A.1.3). The dose (of 8 sessions plus daily exercises) was primarily guided by participant feedback from our previous CART trial, as well as other breathing therapy trials.<sup>31,193,194</sup>
- **D.3.3.2 Fidelity Procedures.** To improve the internal validity of study findings, comprehensive fidelity methods will be implemented. <sup>195</sup> These methods will include standardizing interventionist training and supervision protocols; manualizing CALM Breathing; and monitoring and measuring intervention implementation and

receipt. Intervention fidelity is "the extent to which an intervention's core components have been implemented as planned". 196, p. 377 Two interventionists will be trained and certified by Dr. Norweg to implement CALM Breathing, A 12-hour, standardized training program will be developed consisting of biofeedback demonstrations, case studies, and a mock visit (7 hours); manual assessment techniques (1 hour); and dyspnea, anxiety, behavior change, and MI principles (4 hours). 197,83 Clinicians will implement CALM Breathing. For certification, Dr. Norweg will review recordings and written notes of the first three sessions of CALM Breathing and provide detailed feedback. 198 A random selection of 20% of audio-recorded CALM Breathing intervention sessions and written notes (drawn from different therapy phases)<sup>198</sup> will be audited by Dr. Norweg and discussed during regular supervision meetings to improve interventionists' competence and prevent intervention drift. A fidelity checklist will be used with core CALM Breathing components included. The checklist will use a 0-2 scoring scale and include three domains: session structure, session content, and session tailoring (adapted from another fidelity checklist<sup>199</sup>). For coaching, the Motivational Interviewing Treatment Integrity Scale (MITI-4) will be used, which is well validated and includes four global ratings—Cultivating Change Talk, Softening Sustain Talk, Partnership, and Empathy, with a 1–5 scale. 200-202 CALM Breathing attendance will be tracked closely by the RA. We implemented fidelity monitoring with regular supervision meetings and MITI-4 in our prior CART study.

**D.3.3.3 Wait-List Control Group (Study Phase I).** After referral to CUIMC's PR program, participants randomized to the Wait-List control group will be put on a PR wait list (usual care).

| Table 3. | Table 3. CALM Breathing Sessions. | |
|---|---|---|
| Session | Session Plan | Min |
| 1 | <ul> <li>Introduce CALM Breathing; combine initial interview with capnography assessment; manually evaluate respiratory muscle function and assess for lower ribcage paradox (in supine and sitting).</li> <li>Introduce mind-body connection; educate about role of CO<sub>2</sub>; discuss link between the breath and emotions. Educate about anxiety, and the cycle of breathing and panic, and related physiology. Discuss overall goals, homework, and target goals; train in RR device and exercise log use.</li> </ul> | 40 20 |
| 2–8 | <ul> <li>Review homework exercise log and recorded RR data; problem-solve barriers.</li> <li>Implement tailored CALM Breathing exercises (at rest and with low-moderate intensity) and MI.</li> <li>Collaboratively set target behavior goals and discuss home-based breathing exercises. Borg dyspnea score: max. 4.<sup>77</sup></li> </ul> | 10<br>40<br>10 |

**D.3.3.4 PR Intervention (Standard Care Phase II)**. CUIMC's PR program will be delivered as part of care as usual (**Table 4**). A wait of approximately 6 weeks for PR is typical at New-York Presbyterian / CUIMC

| | Traditional outpatient PR (rolling admission) | CALM Breathing |
|---|---|---|
| Components | Group exercise training (ET) combined with PLB training. <sup>77,203</sup> | Individual interoception-based breathing therapy with capnography <sup>17,72,77</sup> (non-exercise training <sup>204</sup> ). |
| Home Program | Unmonitored walking exercise 1–2 days/week; no biofeedback monitoring. | Monitored home-based breathing exercises; RR biofeedback; goal setting; exercise logging. |
| Coaching | Traditional monitoring and verbal cueing. | Motivational interviewing. |
| Personnel | PT | PT, EP, occupational therapist, or nurse. |
| Frequency | 1-hour sessions, twice per week for 10 weeks. | 1-hour sessions, twice per week for 4 weeks. |
| Exercises | <ul> <li>ET of muscles of ambulation with exercise equipment, such as treadmill or NuStep (30-min), plus 15-min strengthening exercises; O<sub>2</sub> supplementation. No breathing biofeedback.</li> <li>PLB instruction only during exercise training.</li> </ul> | <ul> <li>10 core breathing exercises with ETCO<sub>2</sub> biofeedback in recovery postures at rest and with body movement (gentle stretches and, in later sessions, brief low-moderate intensity PA).</li> <li>Breathing biofeedback (ETCO<sub>2</sub>, RR, airflow pattern).</li> </ul> |
| Education | Verbal and written information. | Education on anxiety; COPD Patient Guide. <sup>205</sup> |

<u>Note</u>: EP = exercise physiologist.  $O_2$  = oxygen. PLB = pursed lips breathing. PT = physical therapist. RR =respiratory rate.

**D.3.4 Study Assessments and Rationale.** Study outcome assessments will be implemented at baseline, 4 weeks (±2 weeks), and at a 3-month follow-up (±2 weeks). Baseline characteristics will include demographics, social history, smoking status, hospitalizations in the last 12 months, medications and supplemental oxygen use, BMI, mMRC, <sup>12</sup> living situation, depression<sup>206</sup>, cognitive deficits, <sup>207</sup> and literacy. <sup>208</sup> All participants will be administered the Mini-International Neuropsychiatric Interview (MINI)<sup>209</sup> by a psychologist to diagnose

psychiatric disorders (anxiety, depression, bipolar disorder, and psychosis). This psychological assessment (not part of standard care) is important to ensure patient eligibility, reduce study risk, and assist with psychological management of participants. All clinical outcome measures are well validated and sensitive to change in COPD or older adults. Medication dosage, intervention doses, and adverse events will be monitored.

#### D.3.4.1 Outcome Measures.

<u>Feasibility (Aim 1):</u> 1) number of participants recruited within 12 months and reasons for excluding patients; 2) drop-out rate and number of participants lost to follow-up; 3) CALM Breathing treatment session attendance rate and homework adherence; 4) fidelity of CALM Breathing implementation; and (5) facilitation of efficient transition to PR (Phase II). [See Study Record and Statistical Design Plan for more information.]<sup>210</sup>

Acceptability (Aim 2): The acceptability of CALM Breathing will be evaluated based on mixed methods data collected from CALM Breathing attendance, drop-out rate, and satisfaction ratings, and from semi-structured interviews. 181,211 Overall satisfaction of CALM Breathing and homework breathing exercises will be evaluated using stand-alone single items from FACIT treatment satisfaction instrument.<sup>211</sup> To assess themes related to satisfaction and addressable challenges, we will conduct 20-30-min semi-structured, in-depth interviews using open-ended questions, either in person or by phone, post-CALM Breathing at 4-weeks and at 3-month followup. 177,212,213 Open-ended questions provide an opportunity for greater understanding of acceptability, satisfaction, and addressable contextual challenges of an intervention, that cannot be elicited from closedended items alone.<sup>214</sup> Participants will be asked a series of open-ended questions developed from our previous qualitative research. 177 To promote honest answers, as much as possible, interviewer will be blinded to patient social status. Those who dropout will also be interviewed and asked about their experiences with the intervention and reasons for dropping out. The interviewer (research assistant, RA) will receive intensive training from Dr. Raveis and Dr. Norweg prior to conducting open-ended interviews. Dr. Raveis will review the transcripts of initial interviews, critique them, and provide feedback before additional interviews are conducted. Throughout the data collection, Dr. Raveis will monitor the data quality by randomly reviewing selected subset of interview transcripts, to assess that the interviewer is continuing to maintain neutrality, facilitating spontaneous flow of material with non-directive and unstructured questions, and using appropriate transitions to move the discussion from one topic to another, while eliciting range, depth and personal context in the interview. Interviews will be audio-recorded and transcribed by the RA. Coders will be separate from the interviewer; and will receive intensive training and supervision from Dr. Raveis. Coders will use coded transcripts. Coded transcripts will be analyzed with Dedoose software. 215 [See SDP for more details on qualitative analyses.]

Secondary Outcome Measures. Clinical: Dyspnea (Chronic Respiratory Disease Questionnaire, CRQ, dyspnea, DMQ-CAT, and modified Borg scale), 22,216,217 anxiety (GAD-7 and Perceived Stress Scale), 218,219 6MWD, 217 PA, 220 ETCO<sub>2</sub> and RR, QOL<sup>221,222</sup>, and lung function<sup>223</sup>, and quality of life (PROMIS SF V20 Social Roles, V10 Fatigue, V10 Sleep Disturbance, V20 Physical Function). PR Utilization/Engagement: We will measure PR uptake, treatment initiation, attrition rate, and patient activation (using the unidimensional 13-item Patient Activation Measure<sup>224,225</sup>), and acceptability of the Massimo Pulse Oximeter (using the "System Usability Scale)".

<u>Mediating (Process) Outcomes</u>: Interoceptive awareness (MAIA scale), <sup>161,226</sup> AS (ASI-16), <sup>227,186</sup> dyspnea self-efficacy, <sup>22</sup> nasal symptoms (SNOT-20), <sup>228</sup> objective sleep (Actigraphy, Sleep Diary and Nonin Wrist Ox2) and depression (PHQ-9). <sup>206,229</sup> [See Study Record and SDP.]

**D.3.5 Statistical Considerations: Feasibility and Acceptability Success Benchmarks (Aims 1 and 2).** Benchmarks were guided by our prior CART study and other studies.<sup>200,230</sup>

**D.3.5.1 Primary Outcome: Feasibility**. We will calculate % and means to determine whether the following success criteria are met; **Table 5**. 32

| Та | Table 5. Feasibility Success Criteria. |
|---|---|
| 1. | 40 participants are recruited within 12 months (±3 months). |
| 2. | ≥75% participant retention at 4-week (±2 week) evaluation and 3-month follow-up. |
| 3. | CALM Breathing session attendance is ≥70%. |
| 4. | CALM Breathing homework exercise adherence is ≥70% for (5 days/week) using RR device data or exercise log. |
| 5. | A mean of 1 is achieved on CALM Breathing fidelity checklist items and mean of 4 on MITI-4 scale. |

- PR intake assessment is scheduled for week 6–10 for ≥75% of all participants.
- **D.3.5.2 Primary Outcome: Acceptability.** Acceptability *a priori* success benchmarks are:  $(1) \ge 70\%$  CALM Breathing attendance; (2) CALM Breathing drop-out rate is  $\le 10-15\%$ ; and (3) mean of  $\ge 2$  "good" satisfaction rating for CALM Breathing treatment overall (item 8 of FACIT; 0-4 scale).  $^{211}$  [See SDP and Study Record].

**D.3.5.3 Secondary Outcomes**. Hypothesis testing will not be conducted for secondary outcomes.

## D.3.6 Challenges and Alternative Strategies.

We have carefully examined the number of potential participants and are confident we have the pool of participants needed. Strategies to ensure participant recruitment efficiency and retention have been carefully considered. Strategies to ensure participant recruitment efficiency and retention have been carefully considered. Strategies to ensure participant recruitment efficiency and retention have been carefully considered. Strategies to ensure participant recruitment efficiency and retention have been carefully considered it was important to include multiple outcomes for improved rigor. To maintain assessor blinding, the RA (not blinded) will evaluate treatment session and homework adherence outcomes that could reveal intervention group allocation. We will use an iterative process to maximize the likelihood of meeting success benchmarks. We considered offering CO<sub>2</sub> biofeedback for home exercises to increase the dose. However, to keep the home program feasible and easy to carry out, we decided to have participants focus on only one biomarker (RR). If the study findings do not support future clinical trials of CALM Breathing, sub-group analyses will be conducted to illuminate the results (e.g., analyzing feasibility by gender or anxiety level). Revisions might then be made to the study eligibility criteria and/or CALM Breathing intervention.

#### D.4 Study Milestones.

| Table 6. R34 MILESTONES (Months 0-24) | Year 1 | | | | Year 2 | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | |
| Aim 1: Evaluate Feasibility of CALM Breathing | | | | | | | | | |
| Start-up: Develop recruitment materials (flyer) and intervention manual; Obtain IRB approval; Develop data management and | Х | Х | | | | | | | |
| tracking systems; Develop manual of procedures (MOP); Hire | | | | | | | | | |
| and train study staff; Establish data safety monitoring board. | | | | | | | | | |
| Ensure timely execution of agreements | Х | Χ | Χ | Χ | Χ | Х | Х | Х | |
| Screen and recruit 40 study participants | | | | 4 | 12 | 12 | 12 | | 40 |
| Complete enrollment/baseline data collection | | | | 4 | 12 | 12 | 12 | | 40 |
| Complete 4-week post-intervention data collection | | | | 4 | 12 | 12 | 12 | | 40 |
| Complete 3-month follow-up data collection | | | | | 4 | 12 | 12 | 12 | 40 |
| Collect primary and secondary endpoints and adverse events | | | | Χ | Χ | Χ | Χ | Χ | |
| Complete treatment fidelity audits | | | | Χ | Χ | Χ | Χ | | |
| Complete data safety/monitoring reports | | Χ | | Χ | | Χ | | Χ | |
| Complete quality control | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | |
| Obtain annual IRB renewal | | | | | Χ | | | Χ | |
| Conduct statistical analyses | | | | Χ | Χ | Χ | Х | Χ | |
| Submit manuscripts to peer-reviewed journals for dissemination | | | | Χ | Χ | Χ | Χ | Χ | |
| Disseminate findings at conferences | | | | | Χ | Χ | Х | Χ | |
| Aim 2: Evaluate Acceptability of CALM Breathing | | | | | | | | | |
| Analyze CALM Breathing acceptability | | | | Χ | Χ | Χ | Χ | Χ | |
| Disseminate findings at conferences and through publications | | | | | Χ | Χ | Χ | Χ | |
| Submit study results to ClinicalTrials.gov | | | | | | | | Χ | |

#### D.5 Study Organization and Research Team.

At Columbia University Irving Medical Center, CALM Breathing will be led by **Dr. Anna Norweg**. Dr. Norweg is an expert in breathing techniques, capnography biofeedback, MI, and behavioral change in COPD. The research team is highly qualified and experienced. At Columbia University, collaborators represent leaders and experts in the fields of rehabilitation (**Dr. Stein**), exercise physiology, COPD, and pulmonary clinical trials (**Dr. DiMango, Dr. Murphy, and Dr. Buchholz**) and neuropsychology (**Dr. Pavol**).

NYU is a subcontract site (IRB study #: i20-00751\_CR1). To complete our study team, we will collaborate with **Dr. Naomi Simon** (who will continue to serve as multiple-PI), **Dr. Oh** (a specialist in biostatistics), and **Dr. Raveis** (a specialist in qualitative analyses). 3-month re-evaluations of 4 already randomized participants occurred at NYU. No new participant recruitment or retention procedures will occur at NYU. The procedures that will occur at NYU include: (1) Dr. Simon will guide and oversee the implementation of the study remotely from NYU via email and Zoom meetings; (2) Dr. Raveis will assist with training the RA in qualitative study procedures and supervise the coding of transcribed interview data remotely via email and Zoom meetings –

transcripts will not include any identifiers; and (3) Dr. Oh will conduct quantitative data analyses for the study using a coded dataset and work closely with the PIs via Zoom and email.

#### D.6 Future, Large-Scale Clinical Trial.

With achievement of clearly established success benchmarks and milestones, we will demonstrate readiness to proceed to implement a large, adequately powered Phase III efficacy trial.<sup>237</sup> The primary hypotheses for the future clinical trial will be that CRQ-dyspnea and 6MWD mean differences will be greater (≥ minimal important differences, MID) in CALM Breathing compared with waitlist control group at 4 weeks. Two primary outcomes of symptom impact are indicated, which have been rated by stakeholders as important.<sup>238</sup> Our Phase III study will have a 12-month follow-up period. We will also explore mechanisms of CALM Breathing.

#### References

- 1. Kochanek KD, Xu J, Murphy SL, Minino AM, Kung HC. Deaths: preliminary data for 2009. *National vital statistics reports: from the Centers for Disease Control and Prevention, National Center for Health Statistics, National Vital Statistics System.* 2011;59(4):1-51.
- 2. Minino AM, Murphy SL, Xu J, Kochanek KD. Deaths: final data for 2008. *National vital statistics reports: from the Centers for Disease Control and Prevention, National Center for Health Statistics, National Vital Statistics System.* 2011;59(10):1-126.
- 3. Solano JP, Gomes B, Higginson IJ. A comparison of symptom prevalence in far advanced cancer, AIDS, heart disease, chronic obstructive pulmonary disease and renal disease. *Journal of pain and symptom management*. 2006;31(1):58-69.
- 4. Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. *Lancet*. 2006;367(9524):1747-1757.
- 5. Ford ES, Murphy LB, Khavjou O, Giles WH, Holt JB, Croft JB. Total and state-specific medical and absenteeism costs of COPD among adults aged >/= 18 years in the United States for 2010 and projections through 2020. *Chest.* 2015;147(1):31-45.
- 6. Mokdad AH, Ballestros K, Echko M, et al. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. *JAMA*: the journal of the American Medical Association. 2018;319(14):1444-1472.
- 7. Khakban A, Sin DD, FitzGerald JM, et al. The Projected Epidemic of COPD Hospitalizations Over the Next 15 Years: A Population Based Perspective. *American journal of respiratory and critical care medicine*. 2016.
- 8. Lopez-Campos JL, Tan W, Soriano JB. Global burden of COPD. Respirology. 2016;21(1):14-23.
- 9. Rabe KF, Hurd S, Anzueto A, et al. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. *American journal of respiratory and critical care medicine*. 2007;176(6):532-555.
- 10. Toy EL, Gallagher KF, Stanley EL, Swensen AR, Duh MS. The economic impact of exacerbations of chronic obstructive pulmonary disease and exacerbation definition: a review. *Copd.* 2010;7(3):214-228.
- 11. Chronic obstructive pulmonary disease among adults--United States, 2011. MMWR Morbidity and mortality weekly report. 2012;61(46):938-943.
- 12. Vogelmeier CF, Criner GJ, Martinez FJ, et al. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. *American journal of respiratory and critical care medicine*. 2017;195(5):557-582.
- 13. Maurer J, Rebbapragada V, Borson S, et al. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. *Chest.* 2008;134(4 Suppl):43s-56s.
- 14. Aliverti A, Kayser B, Macklem PT. A human model of the pathophysiology of chronic obstructive pulmonary disease. *Respirology*. 2007;12(4):478-485.
- 15. Goodwin RD, Scheckner B, Pena L, Feldman JM, Taha F, Lipsitz JD. A 10-year prospective study of respiratory disease and depression and anxiety in adulthood. *Annals of allergy, asthma & immunology : official publication of the American College of Allergy, Asthma, & Immunology.* 2014;113(5):565-570.
- 16. Evans KC, Banzett RB, Adams L, McKay L, Frackowiak RS, Corfield DR. BOLD fMRI identifies limbic, paralimbic, and cerebellar activation during air hunger. *Journal of neurophysiology*. 2002;88(3):1500-1511.
- 17. Paulus MP. The breathing conundrum-interoceptive sensitivity and anxiety. *Depression and anxiety*. 2013;30(4):315-320.
- 18. Parshall MB, Schwartzstein RM, Adams L, et al. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. *American journal of respiratory and critical care medicine*. 2012;185(4):435-452.
- 19. Manning HL, Schwartzstein RM. Pathophysiology of dyspnea. *The New England journal of medicine*. 1995;333(23):1547-1553.
- 20. Mularski RA, Reinke LF, Carrieri-Kohlman V, et al. An official American Thoracic Society workshop report: assessment and palliative management of dyspnea crisis. *Annals of the American Thoracic Society*. 2013;10(5):S98-106.
- 21. Laviolette L, Laveneziana P. Dyspnoea: a multidimensional and multidisciplinary approach. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2014;43(6):1750-1762.

- 22. Norweg A, Ni P, Garshick E, O'Connor G, Wilke K, Jette AM. A multidimensional computer adaptive test approach to dyspnea assessment. *Archives of physical medicine and rehabilitation*. 2011;92(10):1561-1569.
- 23. Cooper CB. The connection between chronic obstructive pulmonary disease symptoms and hyperinflation and its impact on exercise and function. *The American journal of medicine*. 2006;119(10 Suppl 1):21-31.
- 24. Vidotto LS, Carvalho CRF, Harvey A, Jones M. Dysfunctional breathing: what do we know? *Jornal brasileiro de pneumologia : publicacao oficial da Sociedade Brasileira de Pneumologia e Tisilogia.* 2019;45(1):e20170347.
- 25. Law N, Ruane LE, Low K, Hamza K, Bardin PG. Dysfunctional breathing is more frequent in chronic obstructive pulmonary disease than in asthma and in health. *Respiratory physiology & neurobiology.* 2018;247:20-23.
- 26. Boulding R, Stacey R, Niven R, Fowler SJ. Dysfunctional breathing: a review of the literature and proposal for classification. *European respiratory review : an official journal of the European Respiratory Society.* 2016;25(141):287-294.
- 27. Macklem PT. Therapeutic implications of the pathophysiology of COPD. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2010;35(3):676-680.
- 28. Undem BJ, Kollarik M. The role of vagal afferent nerves in chronic obstructive pulmonary disease. *Proceedings of the American Thoracic Society.* 2005;2(4):355-360; discussion 371-352.
- 29. Gardner WN. The pathophysiology of hyperventilation disorders. *Chest.* 1996;109(2):516-534.
- 30. Yang H, Xiang P, Zhang E, et al. Is hypercapnia associated with poor prognosis in chronic obstructive pulmonary disease? A long-term follow-up cohort study. *BMJ open.* 2015;5(12):e008909.
- 31. Ritz T, Rosenfield D, Steele AM, Millard MW, Meuret AE. Controlling asthma by training of Capnometry-Assisted Hypoventilation (CATCH) vs slow breathing: a randomized controlled trial. *Chest.* 2014;146(5):1237-1247.
- 32. Collins EG, Langbein WE, Fehr L, et al. Can ventilation-feedback training augment exercise tolerance in patients with chronic obstructive pulmonary disease? *American journal of respiratory and critical care medicine*. 2008;177(8):844-852.
- 33. Raupach T, Bahr F, Herrmann P, et al. Slow breathing reduces sympathoexcitation in COPD. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2008;32(2):387-392.
- 34. Rocha A, Arbex FF, Sperandio PA, et al. Excess Ventilation in Chronic Obstructive Pulmonary Disease-Heart Failure Overlap. Implications for Dyspnea and Exercise Intolerance. *American journal of respiratory and critical care medicine*. 2017;196(10):1264-1274.
- 35. Ross RM. ATS/ACCP statement on cardiopulmonary exercise testing. *American journal of respiratory and critical care medicine*. 2003;167(10):1451; author reply 1451.
- 36. Weatherald J, Sattler C, Garcia G, Laveneziana P. Ventilatory response to exercise in cardiopulmonary disease: the role of chemosensitivity and dead space. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2018;51(2).
- 37. Nattie E. Julius H. Comroe, Jr., distinguished lecture: central chemoreception: then ... and now. *Journal of applied physiology (Bethesda, Md : 1985).* 2011;110(1):1-8.
- 38. O'Donnell DE, James MD, Milne KM, Neder JA. The Pathophysiology of Dyspnea and Exercise Intolerance in Chronic Obstructive Pulmonary Disease. *Clin Chest Med.* 2019;40(2):343-366.
- 39. Han JN, Stegen K, Simkens K, et al. Unsteadiness of breathing in patients with hyperventilation syndrome and anxiety disorders. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 1997;10(1):167-176.
- 40. Smoller JW, Pollack MH, Otto MW, Rosenbaum JF, Kradin RL. Panic anxiety, dyspnea, and respiratory disease. Theoretical and clinical considerations. *American journal of respiratory and critical care medicine*. 1996;154(1):6-17.
- 41. Laffey JG, Kavanagh BP. Hypocapnia. *The New England journal of medicine*. 2002;347(1):43-53.
- 42. Maddock RJ. The lactic acid response to alkalosis in panic disorder: an integrative review. *The Journal of neuropsychiatry and clinical neurosciences*. 2001;13(1):22-34.
- 43. Friedman SD, Mathis CM, Hayes C, Renshaw P, Dager SR. Brain pH response to hyperventilation in panic disorder: preliminary evidence for altered acid-base regulation. *The American journal of psychiatry*. 2006;163(4):710-715.
- 44. Ritz T. Airway responsiveness to psychological processes in asthma and health. *Frontiers in physiology.* 2012;3:343.

- 45. Weinberger SE, Schwartzstein RM, Weiss JW. Hypercapnia. *The New England journal of medicine*. 1989;321(18):1223-1231.
- 46. Yu L, De Mazancourt M, Hess A, et al. Functional connectivity and information flow of the respiratory neural network in chronic obstructive pulmonary disease. *Human brain mapping*. 2016;37(8):2736-2754.
- 47. Papp LA, Martinez JM, Klein DF, et al. Respiratory psychophysiology of panic disorder: three respiratory challenges in 98 subjects. *The American journal of psychiatry*. 1997;154(11):1557-1565.
- 48. Henningsen P, Gundel H, Kop WJ, et al. Persistent Physical Symptoms as Perceptual Dysregulation: A Neuropsychobehavioral Model and Its Clinical Implications. *Psychosomatic medicine*. 2018;80(5):422-431.
- 49. Kummer F. Panic attacks in COPD and the somato-psycho-somatic feedback. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2010;36(2):457; author reply 457-458.
- 50. Laurin C, Moullec G, Bacon SL, Lavoie KL. Impact of anxiety and depression on chronic obstructive pulmonary disease exacerbation risk. *American journal of respiratory and critical care medicine*. 2012;185(9):918-923.
- 51. Dalal AA, Shah M, Lunacsek O, Hanania NA. Clinical and economic burden of depression/anxiety in chronic obstructive pulmonary disease patients within a managed care population. *Copd.* 2011;8(4):293-299.
- 52. Tsui MS, Lun FC, Cheng LS, et al. Risk factors for hospital readmission for COPD after implementation of the GOLD guidelines. *The international journal of tuberculosis and lung disease : the official journal of the International Union against Tuberculosis and Lung Disease.* 2016;20(3):396-401.
- 53. Atlantis E, Fahey P, Cochrane B, Smith S. Bidirectional associations between clinically relevant depression or anxiety and COPD: a systematic review and meta-analysis. *Chest.* 2013;144(3):766-777.
- 54. Divo M, Cote C, de Torres JP, et al. Comorbidities and risk of mortality in patients with chronic obstructive pulmonary disease. *American journal of respiratory and critical care medicine*. 2012;186(2):155-161.
- 55. O'Donnell DE, Ora J, Webb KA, Laveneziana P, Jensen D. Mechanisms of activity-related dyspnea in pulmonary diseases. *Respiratory physiology & neurobiology*. 2009;167(1):116-132.
- 56. Bouton ME, Mineka S, Barlow DH. A modern learning theory perspective on the etiology of panic disorder. *Psychological review*. 2001;108(1):4-32.
- 57. Simon NM, Weiss AM, Kradin R, et al. The relationship of anxiety disorders, anxiety sensitivity and pulmonary dysfunction with dyspnea-related distress and avoidance. *The Journal of nervous and mental disease*. 2006;194(12):951-957.
- 58. Paulus MP, Stein MB. An insular view of anxiety. Biological psychiatry. 2006;60(4):383-387.
- 59. Stephan KE, Manjaly ZM, Mathys CD, et al. Allostatic Self-efficacy: A Metacognitive Theory of Dyshomeostasis-Induced Fatigue and Depression. *Frontiers in human neuroscience*. 2016;10:550.
- 60. Barrera TL, Grubbs KM, Kunik ME, Teng EJ. A review of cognitive behavioral therapy for panic disorder in patients with chronic obstructive pulmonary disease: the rationale for interoceptive exposure. *Journal of clinical psychology in medical settings.* 2014;21(2):144-154.
- 61. Bandelow B, Baldwin D, Abelli M, et al. Biological markers for anxiety disorders, OCD and PTSD: A consensus statement. Part II: Neurochemistry, neurophysiology and neurocognition. *The world journal of biological psychiatry: the official journal of the World Federation of Societies of Biological Psychiatry.* 2017;18(3):162-214.
- 62. Paulus MP, Stein MB. Interoception in anxiety and depression. *Brain structure & function*. 2010;214(5-6):451-463.
- 63. Van den Bergh O, Zaman J, Bresseleers J, Verhamme P, Van Diest I. Anxiety, pCO2 and cerebral blood flow. International journal of psychophysiology: official journal of the International Organization of Psychophysiology. 2013;89(1):72-77.
- 64. McEwen BS. Stressed or stressed out: what is the difference? *Journal of psychiatry & neuroscience : JPN.* 2005;30(5):315-318.
- 65. Barrett LF, Simmons WK. Interoceptive predictions in the brain. *Nature reviews Neuroscience*. 2015;16(7):419-429.
- 66. Bandelow B, Baldwin D, Abelli M, et al. Biological markers for anxiety disorders, OCD and PTSD a consensus statement. Part I: Neuroimaging and genetics. *The world journal of biological psychiatry : the official journal of the World Federation of Societies of Biological Psychiatry*. 2016;17(5):321-365.
- 67. Sikter A, Rihmer Z, Guevara R. New aspects in the pathomechanism of diseases of civilization, particularly psychosomatic disorders. Part 1. Theoretical background of a hypothesis. *Neuropsychopharmacologia Hungarica* : a Magyar Pszichofarmakologiai Egyesulet lapja = official journal of the Hungarian Association of Psychopharmacology. 2017;19(2):95-105.

- 68. Davenport PW, Vovk A. Cortical and subcortical central neural pathways in respiratory sensations. *Respiratory physiology & neurobiology*. 2009;167(1):72-86.
- 69. Klein DF. False suffocation alarms, spontaneous panics, and related conditions. An integrative hypothesis. *Archives of general psychiatry.* 1993;50(4):306-317.
- 70. Vollmer LL, Strawn JR, Sah R. Acid-base dysregulation and chemosensory mechanisms in panic disorder: a translational update. *Translational psychiatry*. 2015;5:e572.
- 71. Schulz A, Vogele C. Interoception and stress. Frontiers in psychology. 2015;6:1-23.
- 72. Khalsa SS, Adolphs R, Cameron OG, et al. Interoception and Mental Health: A Roadmap. *Biological psychiatry Cognitive neuroscience and neuroimaging*. 2018;3(6):501-513.
- 73. Bordoni B, Marelli F, Bordoni G. A review of analgesic and emotive breathing: a multidisciplinary approach. *Journal of multidisciplinary healthcare*. 2016;9:97-102.
- 74. Stahl JE, Dossett ML, LaJoie AS, et al. Relaxation Response and Resiliency Training and Its Effect on Healthcare Resource Utilization. *PloS one*. 2015;10(10):e0140212.
- 75. Spathis A, Booth S, Moffat C, et al. The Breathing, Thinking, Functioning clinical model: a proposal to facilitate evidence-based breathlessness management in chronic respiratory disease. *NPJ primary care respiratory medicine*. 2017;27(1):27.
- 76. Neuringer A. Operant variability: evidence, functions, and theory. *Psychonomic bulletin & review.* 2002;9(4):672-705.
- 77. Spruit MA, Singh SJ, Garvey C, et al. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. *American journal of respiratory and critical care medicine*. 2013;188(8):e13-64.
- 78. Sikter A, Rihmer Z, Guevara R. New aspects in the pathomechanism of diseases of civilization, particularly psychosomatic disorders. Part 2. Chronic hypocapnia and hypercapnia in the medical practice.

  Neuropsychopharmacologia Hungarica: a Magyar Pszichofarmakologiai Egyesulet lapja = official journal of the Hungarian Association of Psychopharmacology. 2017;19(3):159-169.
- 79. Newman MG, Lafreniere LS, Jacobson NC. Relaxation-induced anxiety: Effects of peak and trajectories of change on treatment outcome for generalized anxiety disorder. *Psychotherapy research : journal of the Society for Psychotherapy Research.* 2018;28(4):616-629.
- 80. Heide FJ, Borkovec TD. Relaxation-induced anxiety: paradoxical anxiety enhancement due to relaxation training. *Journal of consulting and clinical psychology.* 1983;51(2):171-182.
- 81. Rollick SM, WR, Butler, CC. *Motivational interviewing in health care: Helping patients change behavior.* New York: Guilford Press: 2008.
- 82. Rollnick S, Miller WR. What is motivational interviewing? *Behavioural and Cognitive Psychotherapy*. 1995;23:325-334.
- 83. Gutnick D, Reims K, Davis C, Gainforth H, Jay M. Brief action planning to facilitate behavior change and support patient self-management. *Journal of Clinical Outcomes Management*. 2014;21(1):17-29.
- 84. Bandura A. Health promotion by social cognitive means. *Health education & behavior : the official publication of the Society for Public Health Education.* 2004;31(2):143-164.
- 85. Kinzie MB. Instructional design strategies for health behavior change. *Patient Educ Couns.* 2005;56(1):3-15.
- 86. Karasan E, Abid A, Mieloszyk RJ, Krauss BS, Heldt T, Verghese GC. An Enhanced Mechanistic Model For Capnography, With Application To CHF-COPD Discrimination. *Conference proceedings: Annual International Conference of the IEEE Engineering in Medicine and Biology Society IEEE Engineering in Medicine and Biology Society Conference*. 2018;2018:5267-5272.
- 87. Zwerneman K. End-tidal carbon dioxide monitoring: a VITAL sign worth watching. *Critical care nursing clinics of North America*. 2006;18(2):217-225, xi.
- 88. Nagler J, Krauss B. Capnography: a valuable tool for airway management. *Emergency medicine clinics of North America*. 2008;26(4):881-897, vii.
- 89. Siobal MS. Monitoring Exhaled Carbon Dioxide. Respiratory care. 2016;61(10):1397-1416.
- 90. Biedler AE, Wilhelm W, Kreuer S, et al. Accuracy of portable quantitative capnometers and capnographs under prehospital conditions. *The American journal of emergency medicine*. 2003;21(7):520-524.
- 91. Better Physiology.

- 92. Courtney R, Cohen M. Investigating the claims of Konstantin Buteyko, M.D., Ph.D.: the relationship of breath holding time to end tidal CO2 and other proposed measures of dysfunctional breathing. *Journal of alternative and complementary medicine (New York, NY)*. 2008;14(2):115-123.
- 93. Guyton A. Textbook of Medical Physiology. Philadelphia: WB Saunders; 1991.
- 94. Kubota S, Endo Y, Kubota M. Effect of upper torso inclination in Fowler's position on autonomic cardiovascular regulation. *The journal of physiological sciences : JPS.* 2013;63(5):369-376.
- 95. Migliore A. Management of dyspnea guidelines for practice for adults with chronic obstructive pulmonary disease. *Occupational therapy in health care*. 2004;18(3):1-20.
- 96. Nixon RD, Bryant RA. Induced arousal and reexperiencing in acute stress disorder. *Journal of anxiety disorders*. 2005;19(5):587-594.
- 97. Massaroni C, Carraro E, Vianello A, et al. Optoelectronic Plethysmography in Clinical Practice and Research: A Review. *Respiration; international review of thoracic diseases.* 2017;93(5):339-354.
- 98. Okuro RT, Morcillo AM, Ribeiro MA, Sakano E, Conti PB, Ribeiro JD. Mouth breathing and forward head posture: effects on respiratory biomechanics and exercise capacity in children. *Jornal brasileiro de pneumologia : publicacao oficial da Sociedade Brasileira de Pneumologia e Tisilogia*. 2011;37(4):471-479.
- 99. Kim EJ, Choi JH, Kim KW, et al. The impacts of open-mouth breathing on upper airway space in obstructive sleep apnea: 3-D MDCT analysis. European archives of oto-rhino-laryngology: official journal of the European Federation of Oto-Rhino-Laryngological Societies (EUFOS): affiliated with the German Society for Oto-Rhino-Laryngology Head and Neck Surgery. 2011;268(4):533-539.
- 100. Remmers JE. A century of control of breathing. *American journal of respiratory and critical care medicine*. 2005;172(1):6-11.
- 101. Schwarzacher SW, Wilhelm Z, Anders K, Richter DW. The medullary respiratory network in the rat. *The Journal of physiology*. 1991;435:631-644.
- 102. Courtney R, van Dixhoorn J, Cohen M. Evaluation of breathing pattern: comparison of a Manual Assessment of Respiratory Motion (MARM) and respiratory induction plethysmography. *Applied psychophysiology and biofeedback*. 2008;33(2):91-100.
- 103. Ramirez JM. The integrative role of the sigh in psychology, physiology, pathology, and neurobiology. *Progress in brain research.* 2014;209:91-129.
- 104. Grabauskaite A, Baranauskas M, Griskova-Bulanova I. Interoception and gender: What aspects should we pay attention to? *Consciousness and cognition*. 2017;48:129-137.
- 105. Weitzberg E, Lundberg JO. Humming greatly increases nasal nitric oxide. *American journal of respiratory and critical care medicine*. 2002;166(2):144-145.
- 106. de Sa RB, Pessoa MF, Cavalcanti AGL, Campos SL, Amorim C, Dornelas de Andrade A. Immediate effects of respiratory muscle stretching on chest wall kinematics and electromyography in COPD patients. *Respiratory physiology & neurobiology*. 2017;242:1-7.
- 107. Kozlowska K, Walker P, McLean L, Carrive P. Fear and the Defense Cascade: Clinical Implications and Management. *Harvard review of psychiatry*. 2015;23(4):263-287.
- 108. Seth AK, Friston KJ. Active interoceptive inference and the emotional brain. *Philosophical transactions of the Royal Society of London Series B, Biological sciences.* 2016;371(1708).
- 109. Bort-Roig J, Martin M, Puig-Ribera A, et al. Uptake and factors that influence the use of 'sit less, move more' occupational intervention strategies in Spanish office employees. *The international journal of behavioral nutrition and physical activity.* 2014;11:152.
- 110. Watz H, Pitta F, Rochester CL, et al. An official European Respiratory Society statement on physical activity in COPD. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2014;44(6):1521-1537.
- 111. Lahham A, McDonald CF, Mahal A, et al. Acceptability and validity of a home exercise diary used in home-based pulmonary rehabilitation: A secondary analysis of a randomised controlled trial. *The clinical respiratory journal*. 2018;12(6):2057-2064.
- 112. Nilsson LM. Respiration signals from photoplethysmography. *Anesthesia and analgesia*. 2013;117(4):859-865.
- 113. Schoonjans A, Forget P, Labriola L, et al. Pleth variability index combined with passive leg raising-induced pulse pressure variation to detect hypovolemia in spontaneously breathing patients. *Acta anaesthesiologica Belgica*. 2010;61(3):147-150.

- 114. Perel A. Excessive variations in the plethysmographic waveform during spontaneous ventilation: an important sign of upper airway obstruction. *Anesthesia and analgesia*. 2014;119(6):1288-1292.
- 115. Seth AK, Tsakiris M. Being a Beast Machine: The Somatic Basis of Selfhood. *Trends in cognitive sciences*. 2018;22(11):969-981.
- 116. Van den Bergh O, Witthoft M, Petersen S, Brown RJ. Symptoms and the body: Taking the inferential leap. *Neuroscience and biobehavioral reviews.* 2017;74(Pt A):185-203.
- 117. Petzschner FH, Weber LAE, Gard T, Stephan KE. Computational Psychosomatics and Computational Psychiatry: Toward a Joint Framework for Differential Diagnosis. *Biological psychiatry*. 2017;82(6):421-430.
- 118. Overmier JB. Sensitization, conditioning, and learning: can they help us understand somatization and disability? *Scandinavian journal of psychology.* 2002;43(2):105-112.
- 119. Ankawi B, Slepian PM, Himawan LK, France CR. Validation of the Pain Resilience Scale in a Chronic Pain Sample. The journal of pain: official journal of the American Pain Society. 2017.
- 120. Meuret AE, Ritz T, Wilhelm FH, Roth WT, Rosenfield D. Hypoventilation Therapy Alleviates Panic by Repeated Induction of Dyspnea. *Biological psychiatry Cognitive neuroscience and neuroimaging*. 2018;3(6):539-545.
- 121. Craig AD. Interoception: the sense of the physiological condition of the body. *Current opinion in neurobiology.* 2003;13(4):500-505.
- 122. Wadell K, Webb KA, Preston ME, et al. Impact of pulmonary rehabilitation on the major dimensions of dyspnea in COPD. *Copd.* 2013;10(4):425-435.
- 123. Pitta F TT, Spruit MA, Probst VS, Decramer M, Gosselink R. Characteristics of physical activities in daily life in chronic obstructive pulmonary disease. *American journal of respiratory and critical care medicine*. 2005;171:972-977.
- 124. McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. *The Cochrane database of systematic reviews*. 2015(2):Cd003793.
- von Leupoldt A, Taube K, Lehmann K, Fritzsche A, Magnussen H. The impact of anxiety and depression on outcomes of pulmonary rehabilitation in patients with COPD. *Chest.* 2011;140(3):730-736.
- 126. Janssens T, De Peuter S, Stans L, et al. Dyspnea perception in COPD: association between anxiety, dyspnearelated fear, and dyspnea in a pulmonary rehabilitation program. *Chest.* 2011;140(3):618-625.
- 127. Rochester CL, Vogiatzis I, Holland AE, et al. An Official American Thoracic Society/European Respiratory Society Policy Statement: Enhancing Implementation, Use, and Delivery of Pulmonary Rehabilitation. *American journal of respiratory and critical care medicine*. 2015;192(11):1373-1386.
- 128. Mahler DA, Selecky PA, Harrod CG, et al. American College of Chest Physicians consensus statement on the management of dyspnea in patients with advanced lung or heart disease. *Chest*. 2010;137(3):674-691.
- 129. Bruton A, Lee A, Yardley L, et al. Physiotherapy breathing retraining for asthma: a randomised controlled trial. *The Lancet Respiratory medicine*. 2018;6(1):19-28.
- 130. Marciniuk DD, Goodridge D, Hernandez P, et al. Managing dyspnea in patients with advanced chronic obstructive pulmonary disease: a Canadian Thoracic Society clinical practice guideline. *Canadian respiratory journal: journal of the Canadian Thoracic Society.* 2011;18(2):69-78.
- 131. Somfay A, Porszasz J, Lee SM, Casaburi R. Dose-response effect of oxygen on hyperinflation and exercise endurance in nonhypoxaemic COPD patients. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2001;18(1):77-84.
- 132. Eaton T, Garrett JE, Young P, et al. Ambulatory oxygen improves quality of life of COPD patients: a randomised controlled study. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2002;20(2):306-312.
- 133. McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. *The Cochrane database of systematic reviews.* 2015;2:Cd003793.
- 134. King ML. Affordability, accountability, and accessibility in health care reform: implications for cardiovascular and pulmonary rehabilitation. *Journal of cardiopulmonary rehabilitation and prevention*. 2013;33(3):144-152.
- 135. Johnston K, Grimmer-Somers K. Pulmonary rehabilitation: overwhelming evidence but lost in translation? *Physiotherapy Canada Physiotherapie Canada*. 2010;62(4):368-373.
- 136. Cox NS, Oliveira CC, Lahham A, Holland AE. Pulmonary rehabilitation referral and participation are commonly influenced by environment, knowledge, and beliefs about consequences: a systematic review using the Theoretical Domains Framework. *Journal of physiotherapy*. 2017;63(2):84-93.

- 137. Harrison SL, Robertson N, Graham CD, et al. Can we identify patients with different illness schema following an acute exacerbation of COPD: a cluster analysis. *Respiratory medicine*. 2014;108(2):319-328.
- 138. Man WD, Puhan MA, Harrison SL, Jordan RE, Quint JK, Singh SJ. Pulmonary rehabilitation and severe exacerbations of COPD: solution or white elephant? *ERJ open research*. 2015;1(2).
- 139. Jones SE, Green SA, Clark AL, et al. Pulmonary rehabilitation following hospitalisation for acute exacerbation of COPD: referrals, uptake and adherence. *Thorax*. 2014;69(2):181-182.
- 140. Norweg A, Pickard S, Rolle AJ, et al. Anxiety moderates the association of dyspnea with physical function in people with COPD. *American journal of respiratory and critical care medicine*. 2014;189:A2641.
- 141. Bolton CE, Bevan-Smith EF, Blakey JD, et al. British Thoracic Society guideline on pulmonary rehabilitation in adults. *Thorax*. 2013;68 Suppl 2:ii1-30.
- 142. Corner E, Garrod R. Does the addition of non-invasive ventilation during pulmonary rehabilitation in patients with chronic obstructive pulmonary disease augment patient outcome in exercise tolerance? A literature review. *Physiotherapy research international : the journal for researchers and clinicians in physical therapy.* 2010;15(1):5-15.
- 143. Gould RL, Coulson MC, Howard RJ. Efficacy of cognitive behavioral therapy for anxiety disorders in older people: a meta-analysis and meta-regression of randomized controlled trials. *Journal of the American Geriatrics Society*. 2012;60(2):218-229.
- Tolin DF, Billingsley AL, Hallion LS, Diefenbach GJ. Low pre-treatment end-tidal CO2 predicts dropout from cognitive-behavioral therapy for anxiety and related disorders. *Behaviour research and therapy.* 2017;90:32-40.
- 145. Usmani ZA, Carson KV, Heslop K, Esterman AJ, De Soyza A, Smith BJ. Psychological therapies for the treatment of anxiety disorders in chronic obstructive pulmonary disease. *The Cochrane database of systematic reviews*. 2017;3:Cd010673.
- 146. Gendron LM, Nyberg A, Saey D, Maltais F, Lacasse Y. Active mind-body movement therapies as an adjunct to or in comparison with pulmonary rehabilitation for people with chronic obstructive pulmonary disease. *The Cochrane database of systematic reviews.* 2018;10:Cd012290.
- 147. Clarke G, Yarborough BJ. Evaluating the promise of health IT to enhance/expand the reach of mental health services. *General hospital psychiatry*. 2013;35(4):339-344.
- 148. Starcevic V. Reconsidering benzodiazepines in the treatment of panic disorder. *The Australian and New Zealand journal of psychiatry.* 2012;46(3):271-272.
- 149. Lader M. Benzodiazepine harm: how can it be reduced? *British journal of clinical pharmacology.* 2014;77(2):295-301.
- 150. Buffett-Jerrott SE, Stewart SH. Cognitive and sedative effects of benzodiazepine use. *Current pharmaceutical design.* 2002;8(1):45-58.
- 151. Uchida H, Suzuki T, Mamo DC, et al. Benzodiazepine and antidepressant use in elderly patients with anxiety disorders: a survey of 796 outpatients in Japan. *Journal of anxiety disorders*. 2009;23(4):477-481.
- 152. Bandelow B, Sher L, Bunevicius R, et al. Guidelines for the pharmacological treatment of anxiety disorders, obsessive-compulsive disorder and posttraumatic stress disorder in primary care. *International journal of psychiatry in clinical practice*. 2012;16(2):77-84.
- 153. Man WD, Chowdhury F, Taylor RS, et al. Building consensus for provision of breathlessness rehabilitation for patients with chronic obstructive pulmonary disease and chronic heart failure. *Chronic respiratory disease*. 2016;13(3):229-239.
- 154. Kale MS, Federman AD, Krauskopf K, et al. The Association of Health Literacy with Illness and Medication Beliefs among Patients with Chronic Obstructive Pulmonary Disease. *PloS one*. 2015;10(4):e0123937.
- 155. Richardson CR, Franklin B, Moy ML, Jackson EA. Advances in rehabilitation for chronic diseases: improving health outcomes and function. *Bmj.* 2019;365:l2191.
- 156. Jones AW, Taylor A, Gowler H, O'Kelly N, Ghosh S, Bridle C. Systematic review of interventions to improve patient uptake and completion of pulmonary rehabilitation in COPD. *ERJ open research.* 2017;3(1).
- 157. Early F, Wellwood I, Kuhn I, Deaton C, Fuld J. Interventions to increase referral and uptake to pulmonary rehabilitation in people with COPD: a systematic review. *International journal of chronic obstructive pulmonary disease*. 2018;13:3571-3586.
- 158. Ridwan ES, Hadi H, Wu YL, Tsai PS. Effects of Transitional Care on Hospital Readmission and Mortality Rate in Subjects With COPD: A Systematic Review and Meta-Analysis. *Respiratory care*. 2019;64(9):1146-1156.

- 159. Thaler R, Sunstein C. *Nudge: improving decisions about health, wealth, and happiness.* London, England: Penguin Books: 2009.
- 160. Hertwig R, Grune-Yanoff T. Nudging and Boosting: Steering or Empowering Good Decisions. *Perspectives on psychological science : a journal of the Association for Psychological Science*. 2017;12(6):973-986.
- 161. Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). *PloS one*. 2012;7(11):e48230.
- 162. Center PR. Mobile Fact Sheet: who owns cellphones and smartphones. 2019.
- 163. Livermore N, Sharpe L, McKenzie D. Prevention of panic attacks and panic disorder in COPD. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2010;35(3):557-563.
- 164. Sulemanji DS, Bao F, Jiang Y, Kacmarek RM. A unidirectional breathing pattern improves breathing efficiency in subjects with severe COPD. *Respiratory care*. 2014;59(10):1487-1493.
- 165. Barbera JA, Roca J, Ferrer A, et al. Mechanisms of worsening gas exchange during acute exacerbations of chronic obstructive pulmonary disease. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 1997;10(6):1285-1291.
- 166. Bernardi L, Gabutti A, Porta C, Spicuzza L. Slow breathing reduces chemoreflex response to hypoxia and hypercapnia, and increases baroreflex sensitivity. *Journal of hypertension*. 2001;19(12):2221-2229.
- 167. Gorini M, Misuri G, Corrado A, et al. Breathing pattern and carbon dioxide retention in severe chronic obstructive pulmonary disease. *Thorax.* 1996;51(7):677-683.
- 168. Visser FJ, Ramlal S, Dekhuijzen PN, Heijdra YF. Pursed-lips breathing improves inspiratory capacity in chronic obstructive pulmonary disease. *Respiration; international review of thoracic diseases.* 2011;81(5):372-378.
- 169. Roberts SE. The use of pursed lips breathing in stable chronic obstructive pulmonary disease: a systematic review of the evidence. *Physical Therapy Reviews*. 2009;14(4):240-246.
- 170. Davies CD, McGrath PB, Hale LR, Weiner DN, Tolin DF. Mediators of Change in Capnometry Guided Respiratory Intervention for Panic Disorder. *Applied psychophysiology and biofeedback*. 2018.
- 171. Cavalcanti AG, Lima CS, de Sa RB, et al. Influence of posture on the ventilatory pattern and the thoraco-abdominal kinematics of patients with chronic obstructive pulmonary disease (COPD). *Physiotherapy theory and practice*. 2014;30(7):490-494.
- 172. Priori R, Aliverti A, Albuquerque AL, Quaranta M, Albert P, Calverley PM. The effect of posture on asynchronous chest wall movement in COPD. *Journal of applied physiology (Bethesda, Md : 1985).* 2013;114(8):1066-1075.
- 173. Barach AL, Beck GJ. The ventilatory effects of the head-down position in pulmonary emphysema. *The American journal of medicine*. 1954;16(1):55-60.
- 174. Defilippis V, D'Antini D, Cinnella G, Dambrosio M, Schiraldi F, Procacci V. End-tidal arterial CO2 partial pressure gradient in patients with severe hypercapnia undergoing noninvasive ventilation. *Open access emergency medicine : OAEM.* 2013;5:1-7.
- 175. Galia F, Brimioulle S, Bonnier F, et al. Use of maximum end-tidal CO(2) values to improve end-tidal CO(2) monitoring accuracy. *Respiratory care*. 2011;56(3):278-283.
- 176. Norweg A, Whiteson J, Wu Y, et al. Feasibility of Capnography-Assisted Respiratory Therapy in Chronic Obstructive Pulmonary Disease. *Journal of Respiratory and Critical Care Medicine* 2020;201:A6108.
- 177. Norweg A, Kwon S, Whiteson J, et al. Acceptability of Novel Capnography-Assisted Respiratory Therapy in Chronic Obstructive Pulmonary Disease *Journal of Respiratory and Critical Care Medicine* 2020;201:A5508.
- 178. Norweg AM, Whiteson J, Malgady R, Mola A, Rey M. The effectiveness of different combinations of pulmonary rehabilitation program components: a randomized controlled trial. *Chest.* 2005;128(2):663-672.
- 179. Simon NM, Hofmann SG, Rosenfield D, et al. Efficacy of Yoga vs Cognitive Behavioral Therapy vs Stress Education for the Treatment of Generalized Anxiety Disorder: A Randomized Clinical Trial. *JAMA psychiatry.* 2021;78(1):13-20
- 180. Hoge EA, Bui E, Marques L, et al. Randomized controlled trial of mindfulness meditation for generalized anxiety disorder: effects on anxiety and stress reactivity. *The Journal of clinical psychiatry.* 2013;74(8):786-792.
- 181. Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. *International journal of nursing studies*. 2013;50(5):587-592.

- 182. Lewis A, Bruton A, Donovan-Hall M. Uncertainty prior to pulmonary rehabilitation in primary care: A phenomenological qualitative study in patients with chronic obstructive pulmonary disease. *Chronic respiratory disease*. 2014;11(3):173-180.
- 183. Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. *Journal of psychiatric research*. 2011;45(5):626-629.
- 184. Campbell NC, Murray E, Darbyshire J, et al. Designing and evaluating complex interventions to improve health care. *Bmj.* 2007;334(7591):455-459.
- 185. Campbell M, Fitzpatrick R, Haines A, et al. Framework for design and evaluation of complex interventions to improve health. *Bmj.* 2000;321(7262):694-696.
- 186. Vujanovic AA, Arrindell WA, Bernstein A, Norton PJ, Zvolensky MJ. Sixteen-item Anxiety Sensitivity Index: confirmatory factor analytic evidence, internal consistency, and construct validity in a young adult sample from the Netherlands. *Assessment*. 2007;14(2):129-143.
- 187. Matarazzo BB, Brown GK, Stanley B, et al. Predictive Validity of the Columbia-Suicide Severity Rating Scale among a Cohort of At-risk Veterans. *Suicide & life-threatening behavior*. 2018.
- 188. Nasreddine ZS, Phillips NA, Bedirian V, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. *Journal of the American Geriatrics Society.* 2005;53(4):695-699.
- 189. Norweg AW, JH; Veltri, D; Mejia, J; Sweeney, G; Collins, EG; Krishnan, JA; Lu, Y; Haas, F. The effect of music on walk enjoyment and symptoms in adults with chronic lung diseases. . *American journal of respiratory and critical care medicine*. 2019;199:A5732.
- 190. Costello R, Deegan P, Fitzpatrick M, McNicholas WT. Reversible hypercapnia in chronic obstructive pulmonary disease: a distinct pattern of respiratory failure with a favorable prognosis. *The American journal of medicine*. 1997;102(3):239-244.
- 191. Jensen D, Duffin J, Lam YM, et al. Physiological mechanisms of hyperventilation during human pregnancy. *Respiratory physiology & neurobiology*. 2008;161(1):76-86.
- 192. El-Kotob R, Giangregorio LM. Pilot and feasibility studies in exercise, physical activity, or rehabilitation research. *Pilot and feasibility studies*. 2018;4:137.
- 193. Meuret AE, Wilhelm FH, Ritz T, Roth WT. Feedback of end-tidal pCO2 as a therapeutic approach for panic disorder. *Journal of psychiatric research.* 2008;42(7):560-568.
- 194. Deng G, Feinstein MB, Benusis L, Tin AL, Stover DE. Pilot Study of Self-care Breath Training Exercise for Reduction of Chronic Dyspnea. *Journal of cardiopulmonary rehabilitation and prevention*. 2019;39(1):56-59.
- 195. Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. *Clinical psychology review*. 2011;31(1):79-88.
- 196. Nelson MC, Cordray DS, Hulleman CS, Darrow CL, Sommer EC. A procedure for assessing intervention fidelity in experiments testing educational and behavioral interventions. *The journal of behavioral health services & research.* 2012;39(4):374-396.
- 197. Miller WR, Rollnick S. Motivational Interviewing: helping people change. New York, NY: The Guilford Press; 2013.
- 198. Waltz J, Addis ME, Koerner K, Jacobson NS. Testing the integrity of a psychotherapy protocol: assessment of adherence and competence. *Journal of consulting and clinical psychology.* 1993;61(4):620-630.
- 199. Damschroder LJ, Goodrich DE, Kim HM, et al. Development and validation of the ASPIRE-VA coaching fidelity checklist (ACFC): a tool to help ensure delivery of high-quality weight management interventions. *Translational behavioral medicine*. 2016;6(3):369-385.
- 200. Moyers TB, Rowell LN, Manuel JK, Ernst D, Houck JM. The Motivational Interviewing Treatment Integrity Code (MITI 4): Rationale, Preliminary Reliability and Validity. *Journal of substance abuse treatment*. 2016;65:36-42.
- 201. Moyers TB, Martin T, Manuel JK, Hendrickson SM, Miller WR. Assessing competence in the use of motivational interviewing. *Journal of substance abuse treatment*. 2005;28(1):19-26.
- 202. Moyers TB, Manuel JK, Ernst D. Motivational Interviewing Treatment Integrity Coding Manual 4.1. 2014.
- 203. Garvey C, Bayles MP, Hamm LF, et al. Pulmonary Rehabilitation Exercise Prescription in Chronic Obstructive Pulmonary Disease: Review of Selected Guidelines: AN OFFICIAL STATEMENT FROM THE AMERICAN ASSOCIATION OF CARDIOVASCULAR AND PULMONARY REHABILITATION. *Journal of cardiopulmonary rehabilitation and prevention.* 2016;36(2):75-83.
- 204. Nakazawa A, Cox NS, Holland AE. Current best practice in rehabilitation in interstitial lung disease. *Therapeutic advances in respiratory disease*. 2017;11(2):115-128.

- 205. (CHEST) ACoCP. Living Well with COPD: Chronic Bronchitis and Emphysema Your Patient Guide. Glenview, IL: American College of Chest Physicians; 2014: http://www.chestnet.org/Search#q/q=Living%20Well%20with%20COPD.
- 206. Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. *JAMA: the journal of the American Medical Association*. 1999;282(18):1737-1744.
- 207. Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. *Journal of psychiatric research*. 1975;12(3):189-198.
- 208. Morris NS, MacLean CD, Chew LD, Littenberg B. The Single Item Literacy Screener: evaluation of a brief instrument to identify limited reading ability. *BMC family practice*. 2006;7:21.
- 209. Sheehan DV, Lecrubier Y, Sheehan KH, et al. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. *The Journal of clinical psychiatry*. 1998;59 Suppl 20:22-33;quiz 34-57.
- 210. Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. *Archives of internal medicine*. 2006;166(10):1092-1097.
- 211. Peipert JD, Beaumont JL, Bode R, Cella D, Garcia SF, Hahn EA. Development and validation of the functional assessment of chronic illness therapy treatment satisfaction (FACIT TS) measures. *Quality of life research : an international journal of quality of life aspects of treatment, care and rehabilitation.* 2014;23(3):815-824.
- 212. Braun VaC, V. Using thematic analysis in psychology. Qualitative Research in Psychology. 2006;3:77-101.
- 213. Forman J, Heisler M, Damschroder LJ, Kaselitz E, Kerr EA. Development and application of the RE-AIM QuEST mixed methods framework for program evaluation. *Preventive medicine reports*. 2017;6:322-328.
- 214. Dillman DA, Smyth, J. D., Christian, L. M. *Internet, phone, mail, and mixed-mode surveys: the tailored design method.* 4th ed. Hoboken, NJ: John Wiley & Sons; 2014.
- 215. Dedoose. Version 7.0 ed. Los Angeles, CA: SocioCultural Research Consultants, LLC; 2016.
- 216. Schunemann HJ, Griffith L, Jaeschke R, et al. A comparison of the original chronic respiratory questionnaire with a standardized version. *Chest.* 2003;124(4):1421-1429.
- 217. ATS statement: guidelines for the six-minute walk test. *American journal of respiratory and critical care medicine*. 2002;166(1):111-117.
- 218. Wild B, Eckl A, Herzog W, et al. Assessing Generalized Anxiety Disorder in Elderly People Using the GAD-7 and GAD-2 Scales: Results of a Validation Study. *The American journal of geriatric psychiatry : official journal of the American Association for Geriatric Psychiatry*. 2014;22(10):1029-1038.
- 219. Lee EH. Review of the psychometric evidence of the perceived stress scale. *Asian nursing research.* 2012;6(4):121-127.
- 220. Washburn RA, McAuley E, Katula J, Mihalko SL, Boileau RA. The physical activity scale for the elderly (PASE): evidence for validity. *Journal of clinical epidemiology*. 1999;52(7):643-651.
- 221. Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2009;34(3):648-654.
- 222. Lin FJ, Pickard AS, Krishnan JA, et al. Measuring health-related quality of life in chronic obstructive pulmonary disease: properties of the EQ-5D-5L and PROMIS-43 short form. *BMC medical research methodology*. 2014;14:78.
- 223. Culver BH, Graham BL, Coates AL, et al. Recommendations for a Standardized Pulmonary Function Report. An Official American Thoracic Society Technical Statement. *American journal of respiratory and critical care medicine*. 2017;196(11):1463-1472.
- Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. *Health services research*. 2005;40(6 Pt 1):1918-1930.
- 225. Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. *Health services research*. 2004;39(4 Pt 1):1005-1026.
- 226. Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). *PloS one.* 2018;13(12):e0208034.
- 227. Taylor S, Zvolensky MJ, Cox BJ, et al. Robust dimensions of anxiety sensitivity: development and initial validation of the Anxiety Sensitivity Index-3. *Psychol Assess.* 2007;19(2):176-188.

- 228. Piccirillo JF, Merritt MG, Jr., Richards ML. Psychometric and clinimetric validity of the 20-Item Sino-Nasal Outcome Test (SNOT-20). *Otolaryngology--head and neck surgery : official journal of American Academy of Otolaryngology-Head and Neck Surgery*. 2002;126(1):41-47.
- 229. Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. *Journal of general internal medicine*. 2001;16(9):606-613.
- 230. Gallefoss F, Bakke PS. Patient satisfaction with healthcare in asthmatics and patients with COPD before and after patient education. *Respiratory medicine*. 2000;94(11):1057-1064.
- 231. Levkoff S, Sanchez H. Lessons learned about minority recruitment and retention from the Centers on Minority Aging and Health Promotion. *The Gerontologist*. 2003;43(1):18-26.
- 232. Arean PA, Alvidrez J, Nery R, Estes C, Linkins K. Recruitment and retention of older minorities in mental health services research. *The Gerontologist*. 2003;43(1):36-44.
- 233. Yancey AK, Ortega AN, Kumanyika SK. Effective recruitment and retention of minority research participants. *Annual review of public health.* 2006;27:1-28.
- 234. Russell C, Palmer JR, Adams-Campbell LL, Rosenberg L. Follow-up of a large cohort of Black women. *American journal of epidemiology.* 2001;154(9):845-853.
- 235. Guyatt GH, King DR, Feeny DH, Stubbing D, Goldstein RS. Generic and specific measurement of health-related quality of life in a clinical trial of respiratory rehabilitation. *Journal of clinical epidemiology*. 1999;52(3):187-192.
- 236. Early F, Wilson P, Deaton C, et al. Developing an intervention to increase REferral and uptake TO pulmonary REhabilitation in primary care in patients with chronic obstructive pulmonary disease (the REsTORE study): mixed methods study protocol. *BMJ open.* 2019;9(1):e024806.
- 237. Bowen DJ, Kreuter M, Spring B, et al. How we design feasibility studies. *American journal of preventive medicine*. 2009;36(5):452-457.
- 238. Spruit MA, Pitta F, Garvey C, et al. Differences in content and organisational aspects of pulmonary rehabilitation programmes. *The European respiratory journal : official journal of the European Society for Clinical Respiratory Physiology.* 2014;43(5):1326-1337.